# Official Title of Study:

A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Effect of Deucravacitinib on Quality of Life in Participants With Plaque Psoriasis in a Community Setting (ARTISTYK)

NCT Number: NCT05701995

Document Date (Date in which document was last revised): May 25, 2023

Page: 1

Protocol Number: IM011237

Date: 10-May-2022

Revised Date: 25-May-2023

### CLINICAL PROTOCOL IM011237

A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY EVALUATING THE EFFECT OF DEUCRAVACITINIB ON QUALITY OF LIFE IN PARTICIPANTS WITH PLAQUE PSORIASIS IN A COMMUNITY SETTING (ARTISTYK)

Compound: BMS-986165

**Brief Title:** Randomized, double-blind, placebo-controlled study to evaluate the effect of deucravacitinib on quality of life in participants with plaque psoriasis in a community setting

### **Protocol Amendment 02**

Clinical Trial Physician-Medical Monitor Bristol-Myers Squibb Company 86 Morris Ave Summit, NJ 07901

> Teleph<u>one:</u> Email:

Clinical Scientist
Bristol-Myers Squibb Company
3401 Princeton Pike
Lawrenceville, NJ 08648
Telephone:

Email:

### 24-hr Emergency Telephone Number

USA: 1-866-470-2267 International: +1-248-844-7390

# **Bristol-Myers Squibb Company**

Route 206 & Province Line Road Lawrenceville, NJ 08543

Avenue de Finlande 4 B-1420 Braine-l'Alleud, Belgium

### **REGULATORY AGENCY IDENTIFIER NUMBER(S)**

IND: 131,993

NCT: NCT05701995

UTN: U1111-1276-5158

Clinical Protocol BMS-986165

This document is the confidential and proprietary information of Bristol-Myers Squibb Company (BMS) and its global affiliates. By reviewing this document, you agree to keep it confidential and to use and disclose it solely for the purpose of assessing whether your organization will participate in and/or the performance of the proposed BMS sponsored study. Any permitted disclosures will be made only on a confidential "need to know" basis within your organization or to your Independent Ethics Committee(s). Any other use, copying, disclosure or dissemination of this information is strictly prohibited unless expressly authorized in writing by BMS. Any supplemental information (eg, amendments) that may be added to this document is also confidential and proprietary to BMS and must be kept in confidence in the same manner as the contents of this document. Any person who receives this document without due authorization from BMS is requested to return it to BMS or promptly destroy it. References to BMS in this protocol may apply to partners to which BMS has transferred obligations (eg, a Contract Research Organization).

© 2023 Bristol-Myers Squibb Company

# **DOCUMENT HISTORY**

| Document | Date of Issue | Summary of Changes |
|---|---|---|
| Protocol Amendment | 25-May-2023 | The compound number was added to the title page. |
| 02 | | The Sponsor contact information was updated and the Sponsor contact information for the medical monitor was updated . |
| | | • Text was revised to reflect approval of SOTYKTU <sup>TM</sup> (deucravacitinib) in multiple countries at a dose of 6 mg QD. |
| | | • An additional key inclusion criterion was added: moderate-to-severe plaque psoriasis . The text throughout multiple sections was updated accordingly to reflect this change. |
| | | • s-PGA 0/1 at Week 16 was added as a key secondary endpoint and s-PGA assessment was added to the Screening visit. |
| | | • The statistical methods were updated to include a description of the 2 populations of interest (Overall Population and the s-PGA Sub-Population [participants with s-PGA ≥ 3 at baseline]). |
| | | • Added corresponding text on the null hypothesis, definition of estimands, etc for s-PGA 0/1. |
| | | • The following exclusion criterion: "Participants who are not fully vaccinated against SARS-CoV-2 as defined by the local and current national guidelines" was made "Not applicable per Protocol Amendment 02." |
| | | • Additional details were added to clarify guidance for investigators to check and provide counseling to the participants with regard to vaccinations. |

| Document | Date of Issue | Summary of Changes |
|---|---|---|
| | | • The collection of non-serious AEs was removed from Week -2 (Visit 1). |
| | | Details of the external SSC were added. |
| | | <ul> <li>Updated the Schedule of Activities Table to include efficacy assessment of scalp, nail, palmoplantar, inverse, genital, or facial psoriasis at every study visit.</li> </ul> |
| | | Collection of the TSQM was removed from Day 1 (Visit 2) with subsequent change in the endpoint to reflect that the TSQM will be collected starting at Week 4. |
| | | • Added the following footnote to Table 2-2: "The Week 1 visit should not be entered into the IRT system because study intervention is not dispensed at Week 1." |
| | | • Removed 1,25-dihydroxy vitamin D <sub>3</sub> and analogues from the list of exclusionary systemic non-biologic medications. |
| | | The following text: "No concomitant medications (prescription, over-the-counter, or herbal) are to be administered during the study unless prescribed for intervention of specific clinical AEs. Any concomitant therapies must be recorded on the (e)CRF. The investigator should contact and confirm agreement with the Medical Monitor or designee prior to the administration of any concomitant medications." was replaced with: "Concomitant medications (prescription, over the counter, or herbal) should be administered during the study only if they are to be used for treatment of specific medical reasons." |
| | | Additional details were added to clarify which assessments are to be repeated during rescreening. |

| Document | Date of Issue | Summary of Changes |
|---|---|---|
| | | <ul> <li>A row was added to the Schedule of Activities Table to dispense the e-diary device at Screening.</li> <li>A row was added to the Schedule of Activities Table to collect the e-diary device at Week 52.</li> </ul> |
| Protocol Amendment<br>01 | 21-Nov-2022 | <ul> <li>The US FDA approval date was added for the study drug.</li> <li>The duration that participants will wear the wristwatch was increased from 7 days to 14 days before each wear period (ie, prior to Day 1, Week 16, and Week 52).</li> <li>Details about completed and ongoing studies were updated.</li> <li>Pregnant partner surveillance language was removed.</li> <li>Clarifying additions/deletions were made throughout the protocol.</li> <li>Minor administrative changes were made throughout the protocol.</li> </ul> |
| Original Protocol | 19-May-2022 | Not applicable. |

(e)CRF, electronic case report form; AE, adverse event;

FDA, Food and Drug Administration; technology; QD, once daily; SARS-CoV-2, severe acute respiratory syndrome coronavirus 2; s-PGA, static Physician Global Assessment; SSC, Study Steering Committee; TSQM, Treatment Satisfaction Questionnaire for Medication; US, United

States;

# **OVERALL RATIONALE FOR PROTOCOL AMENDMENT 02**

Overall Rationale for Protocol Amendment 02, 25-May-2023

| This protocol has been revised |
|--------------------------------|

Additionally, the rationale for Protocol Amendment 02 was to ensure that the study will enroll participants with moderate-to-severe plaque psoriasis

| SUMMARY OF CHANGES FOR PROTOCOL AMENDMENT 02 | | |
|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Title Page | The compound number was added to the title page. | This change was made to reflect the Sponsor's protocol template. |
| Title Page | The Sponsor contact information was updated and the Sponsor contact information for the medical monitor was updated. | This change was made to reflect changes in the study personnel. |
| Section 1<br>Protocol Summary | Text was revised to reflect approval of SOTYKTU <sup>TM</sup> (deucravacitinib) by | This revision was made to reflect approval of deucravacitinib by |
| Section 3.1<br>Study Rationale | Health Authorities in multiple countries. | Health Authorities in additional countries beyond the US. |
| Section 3.2.1<br>Clinical Development | | |
| Section 6.1 | An additional key inclusion criterion | • |
| Inclusion Criteria | was added: | |
| Section 1 | | |
| Protocol Summary | | |
| Section 3.1 | | |

|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Study Rationale Section 5.1.1 Screening Period Section 5.4 Scientific Rationale for Study Design | The text throughout multiple sections was updated accordingly to reflect this change. | To reflect this additional key inclusion criteria, the text was updated throughout the protocol. |
| Section 2 Schedule of Activities (Table 2-1) | s-PGA assessment was added to the Screening visit. | • |
| Section 1 Protocol Summary Section 4 Objectives and Endpoints (Table 4-1) | s-PGA 0/1 at Week 16 was added as a key secondary endpoint. | |
| Throughout | The text was updated in multiple sections. | The text throughout the protocol was updated to reflect this change. |
| Section 10<br>Statistical Considerations | An additional sub-population was defined for the primary and secondary analyses. Due to additional hypothesis tests within each endpoint using 2 analysis populations, Sample sizes and their corresponding powers are reassessed for each study endpoint for the additional population. | |
| | • The statistical methods were updated to include a description of the 2 populations of interest (Overall Population and the Sub-Population of participants with s-PGA ≥ 3 at baseline). | <ul> <li>To provide additional description of<br/>the analyses that would be<br/>performed for sub-population of<br/>participants with s-PGA ≥ 3 at<br/>baseline.</li> </ul> |
| | • Added corresponding text on the null hypothesis, definition of estimands, etc for s-PGA 0/1. | |
| Throughout | The text was updated in multiple sections. | The text throughout the protocol was updated to reflect this change. |

| Section Number & Title | Description of Change | Brief Rationale |
|---|---|---|
| Section 6.2<br>Exclusion Criteria | • The following exclusion criterion: "Participants who are not fully vaccinated against SARS-CoV-2 as defined by the local and current national guidelines" was made "Not applicable per Protocol Amendment 02." | To minimize barriers for participan<br>enrollment, this exclusion criteria<br>was removed. |
| Section 2 Schedule of Activities (Table 2-1) | Additional details were added to clarify guidance for investigators to check and provide counseling to the participants with regard to vaccinations as follows: Investigators are encouraged to check whether participants have had preventive health measures such as cancer screening (eg, Pap smear, colonoscopy, mammograms) and are up-to-date with recommended vaccinations according to local guidelines (eg, influenza, herpes zoster, SARS-CoV-2). | To clarify and provide guidance for investigators to counsel participants with regard to vaccinations. |
| Section 2 Schedule of Activities (Table 2-2) | | |
| Section 2 Schedule of Activities (Table 2-1) | | |

|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Section 12 | | |
| Section 2 Schedule of Activities (Table 2-1) Section 6.2 Exclusion Criteria | HBV DNA viral load was removed as a required test at screening. | |
| Section 12 Appendices APPENDIX 6 HEPATITIS B VIRUS (HBV) SCREENING | Additionally, a new appendix<br>(APPENDIX 6) providing detailed<br>HBV screening approach was added. | To provide detailed instructions for HBV screening. |
| Section 1 Protocol Summary Section 4 Objectives and Endpoints (Table 4-1) | Similar changes were made to the text describing the safety analyses. | |
| Section 2 Schedule of Activities (Table 2-2) | • The collection of non-serious AEs was removed from Week -2 (Visit 1). | To align with the description in the protocol (Section 9.2.2) which indicates AEs (non-serious) collection begins with the initiation of study treatment. |

|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Section 1 Protocol Summary Section 5.1.6 Data Monitoring Committee and Other Committees | Details of the external SSC were added. | To provide the description and the roles of the SSC in the protocol. |
| Section 2 Schedule of Activities (Table 2-2 and Table 2-3) | Updated the Schedule of Activities<br>Table to include efficacy assessment<br>of scalp, nail, palmoplantar, inverse,<br>genital, or facial psoriasis at every<br>study visit. | In order to be able to capture response and/or potentially disease flare in any of these 'difficult-to-treat' sites throughout the study |
| Section 2 Schedule of Activities (Table 2-2) Section 1 Protocol Summary | Collection of the TSQM was removed<br>from Day 1 (Visit 2) with subsequent<br>change in the endpoint to reflect that<br>the TSQM will be collected starting at<br>Week 4. | TSQM questionnaire was not applicable to be administered prior to the initiation of the IP and was thus removed from Day 1. The TSQM will be collected |
| Section 4 Objectives and Endpoints (Table 4-1) | | starting at Week 4 after the participant has begun treatment. |
| Section 2<br>Schedule of Activities<br>(Table 2-2) | Added the following footnote: "The Week 1 visit should not be entered into the IRT system because study intervention is not dispensed at Week 1." | This revision was made to clarify<br>the IRT system procedures. |
| Section 2<br>Schedule of Activities<br>(Table 2-2 and Table 2-3) | | To have consistent language throughout the protocol. |
| Section 6.2<br>Exclusion Criteria | | |

|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Section 6.2 | | |
| Exclusion Criteria | • Removed 1,25-dihydroxy vitamin D <sub>3</sub> and analogues from the list of exclusionary systemic non-biologic medications. | To reduce participant burden and optimize enrollment this prohibited medication/exclusion criteria was removed. |
| Section 7.7.1 Prohibited and/or Restricted Interventions Section 7.7.2 Permitted Concomitant Medications | • The following text: "No concomitant medications (prescription, over-the-counter, or herbal) are to be administered during the study unless prescribed for intervention of specific clinical AEs. Any concomitant therapies must be recorded on the (e)CRF. The investigator should contact and confirm agreement with the Medical Monitor or designee prior to the administration of any concomitant medications." was replaced with: "Concomitant medications (prescription, over the counter, or herbal) should be administered during the study only if they are to be used for treatment of specific medical reasons." | <ul> <li>This requirement was removed from this Phase 4 study to minimize participant and Investigator burden.</li> <li>Provided clarification to streamline administration and capturing concomitant medications during the study on the eCRF.</li> </ul> |
| Section 6.4.1 Retesting During the Screening Period | Additional details were added to clarify which assessments are to be repeated during rescreening. | To minimize participant burden and optimize enrollment. |
| Section 7.8 Continued Access to Study Intervention After the End of the Study | • The following paragraph was removed: "BMS reserves the right to terminate access to BMS-supplied study intervention if any of the following occur: a) the study is terminated due to safety concerns; b) the development of deucravacitinib is terminated for other reasons, including but not limited to lack of efficacy and/or not meeting the study objectives; c) the participant can obtain medication from a government sponsored or private health program. In all cases BMS will follow local regulations." | This paragraph was not applicable to this Phase 4 study. |

|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Section 2 Schedule of Activities (Table 2-1) | A row was added to the Schedule of<br>Activities Table to dispense the e-<br>diary device at Screening. | To clarify for Investigators that ediary is dispensed at screening. |
| Section 2 Schedule of Activities (Table 2-3) | A row was added to the Schedule of<br>Activities Table to collect the e-diary<br>device at Week 52. | To clarify and remind Investigators<br>that e-diary must be collected at<br>Week 52 visit. |
| All | Minor administrative changes and clarifying edits were made throughout the protocol. | Minor edits were made to improve overall readability, consistency, and to streamline this phase 4 Study protocol following the FDA approval of SOTYKTU <sup>TM</sup> . |

(e)CRF, electronic case report form; AE, adverse event; BMS, Bristol-Myers Squibb Company; COVID-19, coronavirus disease 2019; DNA, deoxyribonucleic acid; FDA, Food and Drug Administration; e-diary, electronic diary;

HBV, hepatis B virus; IB, Investigator's Brochure; IP, investigational product; IRT, interactive response technology; PE, physical examination; QD, once daily; QoL, quality of life; SAE, serious adverse event; SARS-CoV-2, severe acute respiratory syndrome coronavirus 2; s-PGA, static Physician Global Assessment; SSC, Study Steering Committee; TSQM, Treatment Satisfaction Questionnaire for Medication; TYK2, tyrosine kinase 2; US, United States; WHO, World Health Organization.

# **TABLE OF CONTENTS**

| CLINIC | AL PROTOCOL IM011237 | 1 |
|----------------|------------------------------------------------|------------|
| | MENT HISTORY | |
| | LL RATIONALE FOR PROTOCOL AMENDMENT 02 | |
| SUMM | ARY OF CHANGES FOR PROTOCOL AMENDMENT 02 | 6 |
| <b>TABLE</b> | OF CONTENTS | |
| 1 | PROTOCOL SUMMARY | |
| 2 | SCHEDULE OF ACTIVITIES | |
| 3 | INTRODUCTION | |
| 3.1 | Study Rationale | |
| 3.2 | Background | |
| 3.2.1 | Clinical Development | <u></u> 36 |
| | | 36 |
| | | 37 |
| | | 37 |
| | | 38 |
| 1 | OBJECTIVES AND ENDPOINTS | 39 |
| 4<br>5 | STUDY DESIGN | |
| 5.1 | Overall Design | |
| 5.1.1 | Screening Period | |
| 5.1.1 | Intervention Period | |
| 5.1.3 | Week 16 | |
| 5.1.3<br>5.1.4 | Week 20 | |
| 5.1.5 | Week 52 and Safety Follow-up Period | |
| 5.1.6 | Data Monitoring Committee and Other Committees | |
| 5.1.0 | Number of Participants | |
| 5.3 | End of Study Definition | |
| 5.4 | Scientific Rationale for Study Design | |
| J. T | Scientific Rationale for Study Design | |
| 6 | STUDY POPULATION | 45 |
| 6.1 | Inclusion Criteria | |
| 6.2 | Exclusion Criteria | |
| 6.3 | Lifestyle Restrictions | |
| 6.3.1 | Meals and Dietary Restrictions | |
| 6.3.2 | Caffeine, Alcohol and Tobacco | |
| 6.3.3 | Activity | |
| 6.4 | Screen Failures | |
| 6.4.1 | Retesting During the Screening Period | |
| 7 | STUDY INTERVENTION(S) AND CONCOMITANT THERAPY | |
| 7.1 | Study Interventions Administered | |
| 7.2 | Method of Study Intervention Assignment | |
| 7.3 | Blinding | |
| 7.3.1 | Maintaining the Blind | 54 |
| 7.3.2 | Circumstances for Unblinding | |
| 7.4 | Dosage Modification | |

| 7.5 | Preparation/Handling/Storage/Accountability | 55 |
|---|---|---|
| 7.6 | Treatment Compliance | |
| 7.7 | Concomitant Therapy | 56 |
| 7.7.1 | Prohibited and/or Restricted Treatments | 56 |
| <u>7.7.2</u> | Permitted Concomitant Medications | <u></u> 57 |
| | | 58 |
| 7.7.4 | Permitted Vaccines (Including COVID-19 Vaccine) | |
| 7.8 | Continued Access to Study Intervention After the End of the Study | |
| 8 | DISCONTINUATION CRITERIA | |
| 8.1 | Discontinuation From Study Intervention | |
| 8.1.1 | Temporary Discontinuation from Study Intervention | |
| 8.1.2 | Post-Study Intervention Study Follow-up | |
| 8.2 | Discontinuation From the Study | |
| 8.2.1 | Individual Discontinuation Criteria | |
| 8.3 | Lost to Follow-up | |
| 9 | STUDY ASSESSMENTS AND PROCEDURES | |
| 9.1 | Efficacy Assessments | |
| 9.1.1 | Investigator-Administered Assessments | |
| 0.2 | | 65 |
| 9.2 | Adverse Events | |
| 9.2.2 | Time David and Everyone for Collecting AE and SAE before ation | 68 |
| 9.2.2 | Time Period and Frequency for Collecting AE and SAE Information | |
| 9.2.3 | Follow-up of AEs and SAEs | |
| 9.2.4 | Regulatory Reporting Requirements for SAEs | |
| 9.2.5 | PregnancyPregnancy | |
| 9.2.7 | Laboratory Test Result Abnormalities | |
| 9.2.8 | Potential Drug-induced Liver Injury (DILI) | |
| 9.2.9 | Other Safety Considerations | |
| 9.3 | Overdose | |
| 9.4 | Safety | |
| 9.4.1 | Physical Examinations. | |
| 9.4.2 | Vital Signs | |
| 9.4.3 | Electrocardiograms | |
| | | 72 |
| | | 72 |
| | | 74 |
| | | 74 |
| | | 74 |
| | | 74 |
| | | 75 |
| | | 75 |
| | | 75 |
| | | 75 |
| | | 75 |
| 9.10 | Health Economics OR Medical Resource Utilization and Health Economics | 75 |

| 10 | STATISTICAL CONSIDERATIONS | .75 |
|---|---|---|
| 10.1 | Statistical Hypotheses | <u>.</u> 75 |
| | | <i>76</i> |
| | | 77 |
| 10.3 | Analysis Sets | |
| 10.4 | Statistical Analyses | .80 |
| 10.4.1 | General Considerations | .80 |
| 10.4.2 | Primary Endpoint(s) | |
| 10.4.3 | Secondary Endpoint(s) | .84 |
| | | 85 |
| 10.4.5 | Safety Analysis | |
| 10.4.6 | Other Analyses | .85 |
| 10.5 | Interim Analyses | .86 |
| 10.6 | Week 16 Primary Analysis | |
| 11 | REFERENCES | |
| 12 | APPENDICES | |
| <b>APPENDIX</b> | | |
| <b>APPENDIX</b> | | .96 |
| APPENDIX | ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: | |
| | DEFINITIONS AND PROCEDURES FOR RECORDING, | |
| | EVALUATING, FOLLOW-UP, AND REPORTING | 107 |
| | EVENTS | |
| | ON OF SAE1 | |
| | ADVERSE EVENTS1 | |
| | TING AES AND SAES1 | |
| | UP OF AES AND SAES1 | |
| REPORTIN | NG OF SAES TO SPONSOR OR DESIGNEE1 | 110 |
| APPENDIX | | |
| | AND METHODS OF CONTRACEPTION | 111 |
| <b>DEFINITIO</b> | | |
| <b>METHODS</b> | S OF CONTRACEPTION1 | 112 |
| COLLECT | <u>IO</u> N OF PR <u>EGNANCY INFORMATION</u> 1 | 114 |
| | | 115 |
| APPENDIX | | 117 |
| APPENDIX | | |
| | HISTORY | 118 |

### 1 PROTOCOL SUMMARY

### **Protocol Title:**

A MULTICENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY EVALUATING THE EFFECT OF DEUCRAVACITINIB ON QUALITY OF LIFE IN PARTICIPANTS WITH PLAQUE PSORIASIS IN A COMMUNITY SETTING (ARTISTYK)

**Brief Title:** Randomized, double-blind, placebo-controlled study to evaluate the effect of deucravacitinib on quality of life in participants with plaque psoriasis in a community setting

### **Rationale:**

SOTYKTU<sup>TM</sup> (deucravacitinib), a first-in-class, oral, selective, allosteric tyrosine kinase 2 (TYK2) inhibitor is approved in multiple countries for the treatment of adults with moderate-to-severe plaque psoriasis who are candidates for systemic therapy or phototherapy. These approvals were based on the results of the 52-week, randomized, Phase 3, placebo-controlled studies of deucravacitinib 6 mg daily versus placebo and apremilast 30 mg twice daily (BID) (POETYK PSO-1 and PSO-2).

In these 2 Phase 3 studies, in addition to achieving both co-primary clinical efficacy endpoints (Psoriasis Area and Severity Index [PASI] 75 and static Physician Global Assessment [s-PGA] 0/1), deucravacitinib also improved Dermatology Life Quality Index (DLQI) scores. Mean changes from baseline in DLQI were greater for deucravacitinib as early as Week 1 versus placebo in PSO-1 (-3.67 vs -2.18) and PSO-2 (-3.49 vs -2.82) and Week 4 versus apremilast in PSO-1 (-5.63 vs -4.83) and Week 8 in PSO-2 (-7.35 vs -6.31). More deucravacitinib-treated patients achieved  $\geq$  4-point improvement on DLQI meaningful change threshold (MCT  $\geq$  4) at Week 16 versus placebo-treated and apremilast-treated patients in PSO-1 (77.6% vs 43.4% and 68.8%, respectively) and PSO-2 (78.6% vs 44.9% and 69.3%). Similarly, higher responses versus apremilast were maintained through Week 24 in PSO-1 (79.5% vs 67.9%) and PSO-2 (79.2% vs 67.5%). In PSO-1, 81.6% achieved MCT ≥ 4 at Week 52 with continuous deucravacitinib treatment. Results were similar when applying an MCT  $\geq$  5. Higher DLQI 0/1 responses were seen with deucravacitinib vs apremilast and placebo arms at Week 16 in POETYK PSO-1 (40.7% vs 28.6% vs 10.6%) and POETYK PSO-2 (38.0% vs 23.1% vs 9.8%). Better DLQI 0/1 responses were also noted at Week 24 in deucravacitinib vs apremilast in POETYK PSO-1 (47.8% vs 24.2%) and PSO-2 (38.0% vs 23.1%). At Week 52, 46.1% of patients in POETYK PSO-1 maintained their DLQI 0/1 score.





Additionally, this is a US-based study that aims to engage community-based dermatologists to facilitate a more diverse patient enrollment and to assess deucravacitinib in a patient population in a setting more real-world than the Phase 3 clinical trial setting.

# **Objectives and Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To compare the efficacy, as measured by DLQI 0/1, of deucravacitinib versus placebo at Week 16: | DLQI 0/1, defined as proportion of participants achieving DLQI score of 0 or 1 at Week 16 |
| <ul> <li>in participants with plaque psoriasis</li> </ul> | |
| <ul> <li>in the sub-population of participants<br/>with s-PGA ≥ 3 at baseline</li> </ul> | |
| Key Secondary | |
| To compare the efficacy, as measured by<br>reduction from baseline in DLQI, of<br>deucravacitinib versus placebo at Week 16: | <ul> <li>Proportion of participants at Week 16, who achieve a ≥<br/>4-point reduction from baseline in DLQI</li> </ul> |
| <ul> <li>in participants with plaque psoriasis</li> <li>in the sub-population of participants with s-PGA ≥ 3 at baseline</li> </ul> | |
| To compare the efficacy, as measured by<br>whole-body itch NRS score, of deucravacitinib<br>versus placebo at Week 16: | Change from baseline in whole-body itch NRS score at Week 16 |
| <ul> <li>in participants with plaque psoriasis</li> </ul> | |
| o in the sub-population of participants with s-PGA ≥ 3 at baseline | |
| • To compare the efficacy, as measured by s-PGA 0/1, of deucravacitinib versus placebo at Week 16 in the sub-population of participants with s-PGA ≥ 3 at baseline | • s-PGA 0/1 response as a proportion of participants with a s-PGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16 |
| Other Secondary | |
| To assess the safety of deucravacitinib versus<br>placebo in participants with plaque psoriasis<br>between Week 0 and Week 16 | AEs, SAEs, laboratory parameters, and vital signs<br>between Week 0 and Week 16 |

| Objectives | Endpoints |
|---|---|
| AE, adverse event;<br>Index; | DLQI, Dermatology Life Quality NRS, Numerical Rating Scale; |
| | SAE, serious adverse event; |

s-PGA, static Physician Global Assessment;

## **Overall Design:**

This is a Phase 4, multicenter, randomized, double-blind placebo-controlled study comparing the effect of deucravacitinib versus placebo on QoL in patients with moderate-to-severe plaque psoriasis and impaired HRQoL. Participants will undergo screening evaluations within 28 days prior to administration of study intervention to determine eligibility. Following the screening process, approximately 174 participants will be randomized in a 2:1 ratio to either deucravacitinib 6 mg once daily (QD) or placebo, respectively.

It is estimated that approximately 90% of randomized participants (ie, approximately 156 participants) would have baseline s-PGA scores  $\geq$  3.

The duration of study participation is approximately 60 weeks and will be divided into the following periods: screening (up to 4 weeks), treatment (52 weeks), and follow-up (4 weeks).

At Week 16, all participants regardless of their blinded intervention, will be switched to open-label deucravacitinib 6 mg QD bottles through Week 52. Participants and investigators remain blinded to double-blind placebo-controlled period study intervention until the end of the study at Week 52.

Participants will be followed up for safety for 4 additional weeks, from Week 52 through Week 56. Participants who discontinue study intervention early/withdraw prematurely must complete the end of treatment visit. The participant will be asked to return to the clinic to complete the 28-day safety follow-up visit and encouraged to report any serious adverse events or adverse events experienced during this time.

# **Number of Participants:**

It is estimated that approximately 250 enrolled participants will be required to achieve 174 randomized. Approximately 174 participants will be randomized in a 2:1 fashion to deucravacitinib 6 mg QD or placebo matching deucravacitinib QD, respectively.

## **Study Population:**

Men and women  $\geq$  18 years of age diagnosed with stable (defined as no morphology changes or significant flares of disease activity in the opinion of the investigator) moderate-to-severe plaque psoriasis for 6 months or more, and impaired QoL (DLQI score > 5), and who are candidates for phototherapy or systemic therapy will be eligible to participate in the study.

## **Intervention Groups and Duration:**

Participants in both intervention groups will take oral doses of one of the investigational [medicinal] product (IP/IMP), either deucravacitinib or placebo QD, for 16 weeks. At Week 16, all participants, regardless of their blinded intervention, will be switched to open-label deucravacitinib 6 mg QD bottles through Week 52.

## **Study Intervention:**

| Study Intervention for IM011237 | | |
|---|---|---|
| Arm Name | Deucravacitinib<br>(BMS-986165) | Placebo |
| Intervention Name | Deucravacitinib<br>(BMS-986165) | Placebo for deucravacitinib |
| Туре | Drug | Drug |
| Dose Formulation | Tablet | Placebo tablet to match deucravacitinib |
| Unit Dose Strength(s) | 6 mg | n/a |
| Dosage Level(s) | 1 active tablet QD in the morning | 1 placebo tablet QD in the morning |
| Route of Administration | Oral | Oral |
| Use | Experimental | Placebo |
| IMP and NIMP/AxMP | IMP | IMP |
| Sourcing | Provided centrally by the Sponsor | Provided centrally by the Sponsor |
| Packaging and Labeling | Study intervention will be provided in a bottle. Each bottle will be labeled as required per country requirement. | Study intervention will be provided in a bottle. Each bottle will be labeled as per country requirement. |

AxMP, auxiliary medicinal products; IMP, investigational medicinal product; n/a, not applicable; NIMP, non-investigational medicinal product; QD, once daily.

#### **Statistical Methods:**

There are 2 population groups of interest in this study. The Overall Population consists of all participants who were randomized to any treatment arm. The s-PGA  $\geq$  3 Sub-Population consists of all participants who were randomized to any treatment arm in the study with s-PGA  $\geq$  3 at baseline.

The 2 primary hypotheses will be tested simultaneously with a significance level (alpha) of 0.05 (2-sided). If either of the test results is not statistically significant (ie, at least one of null hypotheses is not rejected), then it is deemed that the study objective is not met. Key secondary endpoints will be tested in a hierarchical order only if the primary endpoint achieved statistical significance at the 2-sided 0.05 level on both the Overall Population and the s-PGA  $\geq$  3 Sub-Population. A hierarchical test may proceed to the next key secondary endpoint only if both null hypotheses within a key secondary endpoint are rejected.

The analysis model for the primary efficacy endpoint and secondary binary endpoint will use stratified Cochran-Mantel-Haenszel tests

to compare the response rates of deucravacitinib 6 mg QD to placebo. If expected cell counts are not sufficient for each strata level, then strata levels will be combined for the analysis. Non-responder imputation will be used for binary endpoints for participants who discontinue early or who have otherwise missing endpoint data at the specified timepoint. Sensitivity analyses to be performed for the primary endpoint will be described in the statistical analysis plan.

The analysis model for the continuous secondary endpoint will use analysis of covariance with study intervention

The baseline value will be added into the model as a covariate. Intervention differences based on least-squares means and the corresponding 2-sided 95% confidence intervals will be provided for the difference between deucravacitinib 6 mg QD and placebo.

For the continuous secondary efficacy endpoint, multiple imputation will be used for missing data.

The primary analysis at Week 16 will occur once all randomized participants completed their Week 16 visit or discontinued prior to Week 16. Analyses of the collected efficacy and safety data through Week 16 will be performed. A final analysis will be performed after all participants complete the final safety follow-up visit at Week 56 or post-discontinuation follow-up visit.

IM011237

Deucravacitinib

## **Data Monitoring Committee and Other Committees:**

A Data Monitoring Committee will not be used in the study. This study will use an external Study Steering Committee.

## **Brief Summary:**

The purpose of this study is to evaluate the effect of deucravacitinib on QoL in patients with moderate-to-severe plaque psoriasis. The study will also compare the efficacy and safety of deucravacitinib to placebo in participants with moderate-to-severe plaque psoriasis. This will be a randomized, double-blind placebo-controlled study across multiple centers in a community setting.

The study will compare improvement in QoL in participants treated with deucravacitinib to those treated with placebo during the first 16 weeks. This improvement is defined as DLQI 0/1 score and will be assessed at Week 16. The primary hypotheses are that the odds of achieving DLQI 0/1 score at Week 16 in participants receiving deucravacitinib 6 mg QD are improved compared to participants receiving placebo in both the Overall Population and the s-PGA  $\geq$  3 Sub-Population. In addition, the proportion of participants at Week 16 who achieve a  $\geq$  4-point reduction from baseline in DLQI, the change from baseline in whole-body itch Numerical Rating Scale score at Week 16, and the proportion of participants with s-PGA  $\geq$  3 at baseline who achieve s-PGA 0/1 at Week 16 will also be assessed. Similar assessments for improvement and maintenance of response will be performed at Week 52

The duration of study participation is approximately 60 weeks and will be divided into the following periods: screening (up to 4 weeks), treatment (52 weeks), and follow-up (4 weeks). Following the initial screening study visit, subsequent visits will occur at Week –2, Day 1, Week 1, Week 2, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 40, Week 52, and Week 56.

Participants who have completed the screening procedures and have met the inclusion/exclusion criteria will be randomized on Day 1 in a 2:1 ratio to either deucravacitinib 6 mg QD or placebo, respectively, for the first 16 weeks. At Week 16, all participants, regardless of their blinded intervention, will be switched to open-label deucravacitinib 6 mg QD bottles through Week 52. Participants and investigators will remain blinded to the double-blind study intervention until the end of the study.

## 2 SCHEDULE OF ACTIVITIES

Schedules of activities and procedures are documented in Table 2-1 for the Screening Visit, Table 2-2 for Day -14 and Day 1 through Week 20, and Table 2-3 for Week 24 through Week 52.

**Table 2-1:** Screening Procedural Outline (IM011237)

| Procedure | Screening Visit<br>(-28 Days to -1 Day) | Notes |
|---|---|---|
| Eligibility Assessments | | |
| Informed Consent | X | A participant is considered enrolled only when a protocol-specific informed consent is signed. Must be obtained prior to performing any screening procedures |
| Enroll Participant | X | Obtain number from IRT |
| Inclusion/Exclusion Criteria | X | Includes duration of plaque psoriasis and documentation of presence of plaque psoriasis by the investigator |
| Medical History | X | |
| History of Tobacco Use | X | Include description of current tobacco use (Includes medical marijuana or prescription marijuana taken for medicinal reasons) |
| Psoriasis-related History | X | Includes scalp symptoms, psoriatic arthritis, nail involvement, palmoplantar involvement, genital involvement, inverse psoriasis, history of other forms of psoriasis |
| Psoriasis-related Systemic Treatment | X | History of conventional systemic (eg, methotrexate), biologic, and/or phototherapy. For each therapy, include length of time on treatment and reason(s) for discontinuation (eg, lack of efficacy, intolerance, side effects, loss of access to treatment), if applicable |
| Other Prior and Concomitant Treatments | X | Includes topical treatments and shampoos for psoriasis and all medications for other conditions such as cardiovascular disorders and mood disorder |
| Safety Assessments | | |
| PE | X | Complete PE |

**Table 2-1:** Screening Procedural Outline (IM011237)

| Table 2-1: Screenin | g Procedural Oddine ( | 11/1011237) |
|---|---|---|
| Procedure | Screening Visit<br>(-28 Days to -1 Day) | Notes |
| Physical Measurements | X | Includes height, weight, and BMI |
| Vital Signs | X | Includes (ear or oral) body temperature, respiratory rate, seated blood pressure and heart rate. Blood pressure and heart rate should be measured after the participant has been resting quietly for at least 5 minutes |
| 12-lead ECG | X | 12-lead ECGs should be recorded after the participant has been supine for at least 5 minutes. A single ECG would be collected |
| Laboratory Tests | | |
| Pregnancy Test (Serum) | X | For WOCBP only; see APPENDIX 4. |

**Table 2-1:** Screening Procedural Outline (IM011237)

| Procedure | Screening Visit<br>(-28 Days to -1 Day) | Notes |
|---|---|---|
| | | Serum (minimum sensitivity equivalent units 25 IU/L or equivalent units of hCG) to be done at the Screening Visit. |
| | | The participant must be excluded from participation if the serum pregnancy result is positive. |
| | | If needed to document postmenopausal status, as defined in Section 9.4. |
| FSH | X | Females under the age of 55 years must have a serum FSH level > 40 mIU/mL to confirm menopause. |
| AE Reporting | | |
| Monitor for SAEs | X | All SAEs must be collected from the date of participant's written consent until 30 days post discontinuation of dosing or participant's participation in the study if the last scheduled visit occurs at a later time. All AE (SAEs or nonserious AE) related to SARS-CoV-2 infection collected from time of consent. |
| AE, adverse event; | | BMI, body mass index; |
| ECG, electrocardiogram; | teractive response technologies | FSH, follicle-stimulating hormone; hCG, human chorionic gonadotropin; |
| PE, physical examination; | eractive response teennore | 25.13 |
| SAE, serious adverse eve | | acute respiratory syndrome coronavirus 2;<br>Organization; WOCBP, women of childbearing potential. |

Table 2-2: Day -14 and On-Intervention Procedural Outline (IM011237), Day 1 Through Week 20

| Procedure | Week -2<br>D -14<br>(±1 d)<br>Visit 1 | Day 1<br>Visit 2 | Week 1 D8 (±3 d) Visit 3 | Week 2<br>D15<br>(±3 d)<br>Visit 4 | Week 4<br>D29<br>(±3 d)<br>Visit 5 | Week 8<br>D57<br>(±3 d)<br>Visit 6 | Week 12<br>D85<br>(±3 d)<br>Visit 7 | Week 16<br>D113<br>(±3 d)<br>Visit 8 | Week 20<br>D141<br>(±3 d)<br>Visit 9 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| <b>Eligibility Assessments</b> | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | | X | | | | | | | | |
| Medical History | | X | | | | | | | | |
| Safety Assessments | • | | | | | | | | | |
| Targeted PE | | X | X | X | X | X | X | X | X | |
| Body Weight | | X | | | | | | X | | |
| Vital Signs | X | X | X | X | X | X | X | X | X | |
| Concomitant Medication Use | X | X | X | X | X | X | X | X | X | |
| AE Reporting | | | | | | | | | | |
| Monitor for SAEs | X | X | X | X | X | X | X | X | X | |
| Monitor for Nonserious<br>AEs | | X | X | X | X | X | X | X | X | |

Table 2-2: Day -14 and On-Intervention Procedural Outline (IM011237), Day 1 Through Week 20

| Procedure | Week -2<br>D -14<br>(±1 d) | Day 1<br>Visit 2 | Week 1<br>D8<br>(±3 d) | Week 2<br>D15<br>(±3 d) | Week 4<br>D29<br>(±3 d) | Week 8<br>D57<br>(±3 d) | Week 12<br>D85<br>(±3 d) | Week 16<br>D113<br>(±3 d)<br>Visit 8 | Week 20<br>D141<br>(±3 d)<br>Visit 9 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Tests | Visit 1 | | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | V ISIT O | VISIT | |
| Laboratory Tests | | | | | | | | | | |
| Pregnancy Test (Urine) | | X | | | X | X | X | X | X | WOCBP only |
| <b>Efficacy Assessments</b> | 1 | 1 | | | | | 1 | | | |
| PASI | | X | X | X | X | X | X | X | X | |
| s-PGA | | X | X | X | X | X | X | X | X | |
| ss-PGA | | X | X | X | X | X | X | X | X | |
| PGA-F | | X | X | X | X | X | X | X | X | |
| pp-PGA | | X | X | X | X | X | X | X | X | |
| I-s-PGA | | X | X | X | X | X | X | X | X | |
| s-PGA-G | | X | X | X | X | X | X | X | X | |
| sf-PGA | | X | X | X | X | X | X | X | X | |

Table 2-2: Day -14 and On-Intervention Procedural Outline (IM011237), Day 1 Through Week 20

| Procedure | Week -2<br>D -14 | Day 1<br>Visit 2 | Week 1<br>D8 | Week 2<br>D15 | Week 4<br>D29 | Week 8<br>D57 | Week 12<br>D85 | Week 16<br>D113 | Week 20<br>D141 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| | (±1 d) | V 1510 2 | (±3 d) | (±3 d) | (±3 d) | (±3 d) | (±3 d) | (±3 d) | (±3 d) | |
| | Visit 1 | | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | |
| | <u> </u> | | | | | | | | | |

Table 2-2: Day -14 and On-Intervention Procedural Outline (IM011237), Day 1 Through Week 20

| Procedure | Week -2<br>D -14<br>(±1 d)<br>Visit 1 | Day 1<br>Visit 2 | Week 1 D8 (±3 d) Visit 3 | Week 2<br>D15<br>(±3 d)<br>Visit 4 | Week 4<br>D29<br>(±3 d)<br>Visit 5 | Week 8<br>D57<br>(±3 d)<br>Visit 6 | Week 12<br>D85<br>(±3 d)<br>Visit 7 | Week 16<br>D113<br>(±3 d)<br>Visit 8 | Week 20<br>D141<br>(±3 d)<br>Visit 9 | Notes |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Intervention | | | | | | | | | | |
| Randomization via IRT | | X | | | | | | | | |
| Dispense Study<br>Intervention <sup>a</sup> | | X | | X | X | X | X | X | X | |
| Study Intervention<br>Compliance | | | X | X | X | X | X | X | X | |
| Dispense Wristwatch | X | | | | | | X | | | |
| Collect Wristwatch | | X | | | | | | X | | |
| AE, adverse event;<br>technology; I-s-PGA, Intertri<br>Severity Index; | | | PE, phy | | nation; PG | | | Assessmen | | IRT, interactive response PASI, Psoriasis Area and s; pp-PGA, |

WOCBP, women of childbearing potential;

Note: When multiple assessments are conducted at a single visit, the following is the order in which they should be done as applicable:

1)

Global Assessment;

- 2) Safety assessments (eg, vitals, AEs)
- 3) Clinical efficacy assessments
- 4) Laboratory tests (eg, safety laboratory tests).

<sup>&</sup>lt;sup>a</sup> The Week 1 visit should not be entered into the IRT system because study intervention is not dispensed at Week 1.

Table 2-3: On-Intervention Procedural Outline, (IM011237) Week 24 Through Week 52

| Procedures | Week 24<br>D169<br>(±3 d)<br>Visit 10 | Week 28<br>D197<br>(±3 d)<br>Visit 11 | Week 32<br>D225<br>(±3 d)<br>Visit 12 | Week 40<br>D281<br>(±3 d)<br>Visit 13 | Week 52<br>(EOT or ET <sup>a</sup> )<br>D365<br>(±3 d)<br>Visit 14 | Safety Follow-up<br>(Week 56 or<br>Post-Treatment<br>Follow up <sup>a</sup> )<br>D393<br>(±3 d)<br>Visit 15 | Notes |
|---|---|---|---|---|---|---|---|
| Safety Assessments | | | | | _ | | |
| Complete PE | | | | | X | X | |
| Targeted PE | X | X | X | X | | | |
| Body Weight | | | | | X | X | |
| Vital Signs | X | X | X | X | X | X | |
| Concomitant Medication Use | X | X | X | X | X | X | |
| AE Reporting | | | | | | | |
| Monitor for AEs and SAEs | X | X | X | X | X | X | |
| Pregnancy Test (Urine) | X | X | X | X | X | X | WOCBP only |
| Clinical Efficacy Assessments | V | V | V | V | V | | |
| PASI | X | X | X | X | X | | |
| BSA | X | X | X | X | X | | |
| s-PGA | X | X | X | X | X | | |
| ss-PGA | X | X | X | X | X | | |
| PGA-F | X | X | X | X | X | | |

Table 2-3: On-Intervention Procedural Outline, (IM011237) Week 24 Through Week 52

| Procedures | Week 24<br>D169<br>(±3 d)<br>Visit 10 | Week 28<br>D197<br>(±3 d)<br>Visit 11 | Week 32<br>D225<br>(±3 d)<br>Visit 12 | Week 40<br>D281<br>(±3 d)<br>Visit 13 | Week 52<br>(EOT or ET <sup>a</sup> )<br>D365<br>(±3 d)<br>Visit 14 | Safety Follow-up<br>(Week 56 or<br>Post-Treatment<br>Follow up <sup>a</sup> )<br>D393<br>(±3 d)<br>Visit 15 | Notes |
|---|---|---|---|---|---|---|---|
| pp-PGA | X | X | X | X | X | | |
| I-s-PGA | X | X | X | X | X | | |
| s-PGA-G | X | X | X | X | X | | |
| sf-PGA | X | X | X | X | X | | |

Table 2-3: On-Intervention Procedural Outline, (IM011237) Week 24 Through Week 52

| Procedures | Week 24<br>D169<br>(±3 d)<br>Visit 10 | Week 28<br>D197<br>(±3 d)<br>Visit 11 | Week 32<br>D225<br>(±3 d)<br>Visit 12 | Week 40<br>D281<br>(±3 d)<br>Visit 13 | Week 52<br>(EOT or ET <sup>a</sup> )<br>D365<br>(±3 d)<br>Visit 14 | Safety Follow-up<br>(Week 56 or<br>Post-Treatment<br>Follow up <sup>a</sup> )<br>D393<br>(±3 d)<br>Visit 15 | Notes |
|---|---|---|---|---|---|---|---|
| Study Intervention | | | | | | | |
| Dispense Study Intervention | X | X | X | X | | | |
| Study Intervention Compliance | X | X | X | X | X | | |
| Dispense Wristwatch | | | | X | | | |
| Collect Wristwatch | | | | | X | | |
| Collect e-diary | | | | | X | | |
| AE, adverse event; BSA, body surface area; d, da EOT, end of treatment; ET, early termination; I-s- PASI, Psoriasis Area and Severity Index; Physician Global Assessment; SAE, serio Face; s-PGA, static Physician Global Assessment; | PGA, Intertrigues | ent; | PE, 1 | ohysical exar | sf-PGA, s | igational product; Physician Global Asse pp tatic Physician Globalss-PGA, scalp-specifi | -PGA, palmoplantar |

<sup>&</sup>lt;sup>a</sup> EOT/ET visit for participants who discontinue treatment any time prior to completing Week 52 of active treatment period. Safety follow-up visit occurs 28 days ± 3 days after the last dose of study treatment.

Note: When multiple assessments are conducted at a single visit, the following is the order in which they should be done as applicable:

- 1)
- 2) Safety assessments (eg, vitals, AEs)
- 3) Clinical efficacy assessments
- 4) Laboratory tests (eg, safety laboratory tests).

#### 3 INTRODUCTION

### **Plaque Psoriasis**

Psoriasis is a chronic inflammatory disorder, characterized primarily by erythematous scaly plaques, that affects up to 3% of the general population. Men and women are equally affected, and it can present at any age. <sup>1,2</sup> Several studies have observed a bimodal distribution of psoriasis onset with the first peak ranging from 15 to 22 years of age, and the second peak ranging from 55 to 60 years of age. <sup>3,4,5</sup> The most common form of psoriasis (58% to 97%) is plaque psoriasis (psoriasis vulgaris), with less common variants being guttate, pustular, inverse (flexural), and erythrodermic psoriasis. The disease can have a fluctuating relapsing course, with flares that may be induced by factors such as infections, trauma, smoking, and stress.<sup>3</sup> Psoriasis can involve skin in any part of the body; particularly disabling is the involvement of specific anatomic regions, such as hands and feet (palmoplantar), face, scalp, genital, and nails. Psoriasis has been associated with major changes in patients' psychosocial, emotional, and physical functioning. Psoriasis may impact patients' lives as much or more than other major medical conditions. These may include psychological stress, embarrassment, stigma, and physical discomfort, which are not reflected in objective measures of skin disease severity (Psoriasis Area Severity Index [PASI], body surface area [BSA], static Physician Global Assessment [s-PGA]). Over time, these may result in significant worsening in overall emotional well-being, social functioning, productivity at work or school, self-care activities and self-esteem may worsen. Furthermore, the quality of life (QoL) of patients with psoriasis affecting sensitive areas may be disproportionately impacted relative to the affected area. For example, the presence of lesions in highly visible areas can affect a patient's self-esteem, whereas involvement of the palms can make activities of daily living challenging. Nail or hand psoriasis can be a financial burden due to reduced workplace productivity. Scalp psoriasis is frequently associated with pain, itching, and bleeding, and is associated with a disproportionate impact on QoL and psychosocial impairment.<sup>6</sup>

Clinician-reported outcomes for disease severity (PASI, BSA, and s-PGA) may not adequately capture patients' lived experience of the disease. Patient-reported outcome (PRO) measures may provide complementary information, allowing clinicians to better understand the patient's unique experience of living with psoriasis, which could facilitate individualized treatment. Evaluating patients with clinician-reported outcomes (BSA or PASI) or PRO measures alone could lead to an incomplete understanding of disease severity, which may lead to undertreatment or overtreatment.<sup>7,8,9</sup>

Importantly, correlation between Dermatology Life Quality Index (DLQI), which is a standard tool to assess the impact of psoriasis on patients' QoL in clinical studies, and PASI in patients with BSA < 10% has not been fully determined. Furthermore, the National Psoriasis Foundation survey (2003 to 2011) revealed that 30% of patients with 3% to 10% BSA received treatment solely with topical medications and 24% to 36% of psoriasis patients felt that they were untreated. Many patients with BSA < 10% (range: 7.1% to 8.4%) report a large impact on their QoL (DLQI range: 10.2 to 12.2).  $^{10,11}$ 

Treatments for psoriasis include topical preparations (eg, corticosteroids, vitamin D analogues, calcineurin inhibitors, salicylic acid, urea, and coal tar); phototherapy modalities, including broad-band and narrow-band ultraviolet (UV)B; and systemic therapies. In moderate-to-severe disease, systemic treatments are usually needed and may include oral agents (retinoids, methotrexate, cyclosporine, and apremilast) or injectables (eg, biologics such as tumor necrosis factor [TNF] inhibitors etanercept, infliximab, and adalimumab) anti–interleukin [IL]-12/23p40 antibody [ustekinumab], IL-17 antagonists [secukinumab, ixekizumab, and brodalumab], and anti–IL-23p19 antibody [guselkumab, tildrakizumab and risankizumab]. Many of these treatments are associated with increased risk of adverse events (AEs) such as hepatotoxicity and neutropenia (methotrexate); 12 nephrotoxicity (cyclosporine); 13 depression and weight loss (apremilast); 14 serious infections (cytokine inhibitors); 15,16,17,18 and candidiasis and Crohn's disease (IL-17 antagonists). 18,19,20

Although effective therapeutic options are available, undertreatment or nontreatment of psoriasis has been reported in up to half of surveyed patients (based on absence of treatment and/or dissatisfaction with treatment). Many patients with moderate-to-severe disease are still being managed with only topicals, and many patients consider their psoriasis treatment to be inadequate. Accordingly, there remains a need for more effective oral options, when compared with currently available agents, that would improve efficacy responses, increase adherence to treatment and improve various domains of patients' QoL.

# 3.1 Study Rationale

SOTYKTU<sup>TM</sup> (deucravacitinib), a first-in-class, oral, selective, allosteric tyrosine kinase 2 (TYK2) inhibitor is approved in multiple countries for the treatment of adults with moderate-to-severe plaque psoriasis who are candidates for systemic therapy or phototherapy. These approvals were based on the results of completed 52-week, randomized, Phase 3, placebo-controlled studies of deucravacitinib 6 mg daily (BMS-986165) versus placebo and apremilast 30 mg twice daily (BID) (POETYK PSO-1 and PSO-2).

In these 2 Phase 3 studies, in addition to achieving both co-primary clinical efficacy endpoints (PASI 75 and s-PGA 0/1), deucravacitinib also improved DLQI scores. Mean changes from baseline in DLQI were greater for deucravacitinib as early as Week 1 versus placebo in PSO-1 (-3.67 vs -2.18) and PSO-2 (-3.49 vs -2.82) and Week 4 versus apremilast in PSO-1 (-5.63 vs -4.83) and Week 8 in PSO-2 (-7.35 vs -6.31). More deucravacitinib-treated patients achieved  $\geq$  4-point improvement on DLQI meaningful change threshold (MCT  $\geq$  4) at Week 16 versus placebo-treated and apremilast-treated patients in PSO-1 (77.6% vs 43.4% and 68.8%, respectively) and PSO-2 (78.6% vs 44.9% and 69.3%). Similarly, higher responses versus apremilast were maintained through Week 24 in PSO-1 (79.5% vs 67.9%) and PSO-2 (79.2% vs 67.5%). In PSO-1, 81.6% achieved MCT  $\geq$  4 at Week 52 with continuous deucravacitinib treatment. Results were similar when applying an MCT  $\geq$  5. Higher DLQI 0/1 responses were seen with deucravacitinib vs apremilast and placebo arms at Week 16 in POETYK PSO-1 (40.7% vs 28.6% vs 10.6%) and POETYK PSO-2 (38.0% vs 23.1% vs 9.8%). Better DLQI 0/1 responses were also noted at Week 24 in deucravacitinib vs apremilast in POETYK PSO-1 (47.8% vs 24.2%)

and PSO-2 (38.0% vs 23.1%). At Week 52, 46.1% of patients in POETYK PSO-1 maintained their DLQI 0/1 score.



Additionally, this is a US-based study that aims to engage community-based dermatologists to facilitate a more diverse patient enrollment and to provide a more real-world patient population than was studied in Phase 3 studies.

# 3.2 Background

TYK2 is a nonreceptor tyrosine kinase associated with receptors for the p40-containing cytokines IL-12 and IL-23, as well as the Type I interferon (IFN) receptor, and is required for the activation of their downstream signaling pathways. TYK2 catalyzes the phosphorylation of the intracellular receptor domains and signal transducer and activator of transcription (STAT) proteins resulting in the activation of STAT-dependent transcription and functional responses specific for these cytokines. PEC, 22,23,24 Because TYK2-dependent cytokines (eg, Type I IFNs, IL-12, IL-23) are distinct from those dependent on closely related Janus kinase (JAK) family members JAK1/JAK3 (eg, IL-2, IL-15, IL-7) or JAK2 (eg, erythropoietin, thrombopoietin, GM-CSF), a TYK2 inhibitor would be expected to have a distinctly different effects than inhibitors of other JAK family kinases. TYK2-dependent pathways and the cytokine networks they modulate (eg, IL-23/IL-17, IFNα) have been implicated in the pathophysiology of multiple immune-mediated diseases, including psoriasis, lupus, spondylarthritis, and Crohn's disease.

Deucravacitinib is a potent, highly selective, oral, small molecule inhibitor of TYK2. A comprehensive in vitro and in vivo characterization of deucravacitinib has been established and supports the development of this compound in humans. Inhibition of TYK2 is expected to provide therapeutic benefit for participants with psoriasis for multiple reasons: 1) Many of the pathways
in the TYK2 signaling cascade (IL-23 and the downstream mediators IL-17 and IL-22; IFN $\alpha$ ) are involved in the pathogenesis of psoriasis. <sup>21</sup> 2) Biologic agents targeting the IL-17, IL-23p19, and IL-12/23 p40 pathways have been approved for and are highly efficacious in the treatment of psoriasis.

A detailed description of the chemistry, pharmacology, efficacy, and safety of deucravacitinib is provided in the Investigator's Brochure (IB).<sup>26</sup>

#### 3.2.1 Clinical Development

The clinical development program for deucravacitinib consists of multiple studies in healthy volunteers, participants with renal or hepatic insufficiency, and participants with psoriasis, alopecia areata, psoriatic arthritis, systemic lupus erythematosus, lupus nephritis, Crohn's disease, and ulcerative colitis.

In adult participants with moderate-to-severe psoriasis, 1 Phase 2 study (IM011011) and 2 Phase 3 studies (IM011046 and IM011047) have been completed. Study IM011011 was a 12-week, randomized, placebo-controlled study conducted with 5 deucravacitinib intervention arms ranging from 3 mg every other day to 12 mg once daily (QD). Studies IM011046 and IM011047 were pivotal, double-blind, placebo- and active-controlled 52-week, Phase 3 studies. Based on these studies, SOTYKTU<sup>TM</sup> (deucravacitinib), a first-in-class, oral, selective, allosteric TYK2 inhibitor was approved in multiple countries for the treatment of adults with moderate-to-severe plaque psoriasis who are candidates for systemic therapy or phototherapy.

There are 2 other completed Phase 3 studies for adult participants with moderate-to-severe plaque psoriasis (IM011065 and IM011066) and an ongoing long-term extension study (IM011075). IM011065 is a double-blind, placebo-controlled, 52-week study conducted in China, Singapore, South Korea, and Taiwan; IM011066 is a single-arm, open-label study conducted in Japan; IM011075 is an open-label study to evaluate the long-term safety, tolerability, and efficacy of deucravacitinib in participants with psoriasis who were previously enrolled in an applicable parent study (IM011046, IM011047, IM011065, or IM011066).

The clinical pharmacology profile of deucravacitinib has been characterized based on the results of multiple clinical pharmacology studies as well as population pharmacokinetics (PK) and exposure-response analyses that incorporated data from Phase 1, Phase 2, and Phase 3 studies in adult participants with moderate-to-severe psoriasis.

A detailed description is provided in the deucravacitinib IB.<sup>26</sup>







# 4 OBJECTIVES AND ENDPOINTS

Table 4-1: Objectives and Endpoints

| | Objectives | Endacinta | |
|---|---|---|---|
| _ | Objectives | | Endpoints |
| Pri | Primary | | |
| • | To compare the efficacy, as measured by DLQI 0/1, of deucravacitinib versus placebo at Week 16: o in participants with plaque psoriasis o in the sub-population of participants with s-PGA ≥ 3 at baseline | • | DLQI 0/1, defined as proportion of participants achieving DLQI score of 0 or 1 at Week 16 |
| Ke | y Secondary | | |
| • | To compare the efficacy, as measured by reduction from baseline in DLQI, of deucravacitinib versus placebo at Week 16: o in participants with plaque psoriasis o in the sub-population of participants with s-PGA ≥ 3 at baseline | • | Proportion of participants at Week 16, who achieve a ≥ 4-point reduction from baseline in DLQI |
| • | To compare the efficacy, as measured by whole-body itch NRS score, of deucravacitinib versus placebo at Week 16: o in participants with plaque psoriasis o in the sub-population of participants with s-PGA $\geq$ 3 at baseline | • | Change from baseline in whole-body itch NRS score at Week 16 |
| • | To compare the efficacy, as measured by s-PGA $0/1$ , of deucravacitinib versus placebo at Week 16 in the sub-population of participants with s-PGA $\geq 3$ at baseline | • | s-PGA 0/1 response as a proportion of participants with a s-PGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16 |
| Other Secondary | | | |
| • | To assess the safety of deucravacitinib versus placebo in participants with plaque psoriasis between Week 0 and Week 16 | • | AEs, SAEs, laboratory parameters, and vital signs between Week 0 and Week 16 |

Table 4-1: Objectives and Endpoints



## 5 STUDY DESIGN

## 5.1 Overall Design

This study (IM011237) is a Phase 4, multicenter, randomized, double-blind, placebo-controlled study to evaluate the effect of deucravacitinib on QoL in patients with plaque psoriasis and impaired HRQoL. A total of approximately 174 qualified participants with moderate-to-severe

plaque psoriasis will be randomized. It is estimated that approximately 90% of randomized participants (ie, approximately 156 participants) would have baseline s-PGA scores  $\geq 3$ .

The duration of study participation is approximately 60 weeks and will be divided into the following periods: screening (up to 4 weeks), intervention (52 weeks), and safety follow-up (4 weeks).

Physical examination (PE), clinical laboratory evaluations, and other assessments will be done at select visits during the study. Participants in this study will be monitored for AEs.

## 5.1.1 Screening Period

Participants will be evaluated during the screening period (up to 4 weeks/28 days) to ensure they meet eligibility criteria. A detailed medical history will be done at this time, as well as a complete PE. Psoriasis-related history, which will include length of diagnosis, s-PGA score, DLQI score, and history of systemic intervention will be assessed at Screening.

If a participant exceeds the 28-day screening period due to a study-related procedure (eg, waiting for a study-related laboratory value), the participant must be reconsented. A new participant identification number will be assigned by interactive response technology (IRT) at the time of re-enrollment. In this situation, the fewest number of procedures from the initial screening should be repeated to qualify the participant, while maintaining participant safety and eligibility. In these cases, the site should consult with the BMS Medical Monitor (or designee).

#### 5.1.2 Intervention Period

Participants who have completed the screening procedures and have met the inclusion/exclusion criteria will be randomized on Day 1 in a 2:1 ratio to either deucravacitinib 6 mg QD or placebo, respectively.

Dummy tablets (placebo to deucravacitinib 6 mg tablets) will be administered to participants to maintain blinding (Section 7.1).

All participants will receive a wristwatch to monitor sleep quality for 14 days prior to Day 1 to be worn for 14 days. This wristwatch will be returned to the study site on Day 1 as listed in the Schedule of Activities (Section 2). This wristwatch will be returned to all participants again on Weeks 12 and 40 to be worn for 14 days prior to Week 16 and Week 52 and will be returned to the study sites as per the Schedule of Activities (Section 2).

#### 5.1.3 Week 16

All efficacy endpoints and safety will be assessed at Week 16. At Week 16, all participants, regardless of their blinded intervention, will be switched to open-label deucravacitinib 6 mg QD bottles through Week 52. All participants will return their wristwatches at the Week 16 visit.

#### 5.1.4 Week 20

#### 5.1.5 Week 52 and Safety Follow-up Period

The safety follow-up period is a 28-day window after the Week 52 visit. The participant will be encouraged to report any SAEs or AEs experienced during this time.

The end of treatment (EOT) visit will be completed for participants who discontinue study intervention early. The participant will be asked to return to the clinic to complete the 28-day safety follow-up visit.

All participants will return their wristwatches at the Week 52 visit.

The study design schematic is presented in Figure 5.1.5-1.

Figure 5.1.5-1: Study Design Schema



PBO, placebo; QD, once daily.

#### 5.1.6 Data Monitoring Committee and Other Committees

A Data Monitoring Committee will not be used in the study.

Other Committee Charters will describe the procedures related to the committee operations in greater detail.

## 5.1.6.1 External Study Steering Committee (SSC)

The SSC is a committee composed of external experts who assist with the study strategy, protocol development, site identification and patient recruitment strategies. The SSC responsibilities, authorities, and procedures will be documented and followed according to the SSC Charter.

#### 5.2 Number of Participants

It is estimated that approximately 250 enrolled participants will be required to achieve 174 randomized. Approximately 174 participants will be randomized in a 2:1 fashion to deucravacitinib 6 mg QD or placebo matching deucravacitinib QD, respectively.

It is estimated that approximately 90% of randomized participants (ie, approximately 156 participants) would have baseline s-PGA scores  $\geq 3$ .

## 5.3 End of Study Definition

The duration of study participation for individual participants is expected to be up to 60 weeks (420 days), which includes screening (up to 4 weeks), intervention (52 weeks) and follow-up (4 weeks) periods.

The start of the study is defined as the first visit for the first participant screened.

The end of study is defined as the last participant last visit or scheduled procedure shown in the Schedule of Activities (Section 2) for the last participant.

Study completion is defined as the final date on which data were or is expected to be collected if this is not the same.

# 5.4 Scientific Rationale for Study Design

This Phase 4 study will be conducted in a population of participants with stable moderate-to-severe plaque psoriasis who are candidates for systemic psoriasis therapy. Additional key inclusion criterion is DLQI score > 5, which captures participants with moderate-to-severe impact on HRQoL. The study is designed to compare the efficacy of deucravacitinib to placebo in achieving DLQI 0/1 at Week 16. DLQI 0/1 is a standard measure in clinical studies of demonstrating efficacy of systemic psoriasis treatments on QoL. Additional analyses, including formal statistical hypothesis testing, will also be performed in the participant sub-population with s-PGA  $\geq 3$  at baseline for s-PGA 0/1 response at Week 16

s-PGA 0/1 is a standard measure in clinical trials of demonstrating efficacy of systemic psoriasis interventions. A placebo arm is included in this study for a short duration of 16 weeks to provide a control for the natural fluctuation of psoriasis activity that may occur and to provide a safety standard for comparison. Participants in the placebo arm will be switched to deucravacitinib at Week 16 to provide them psoriasis treatment after the endpoints are collected. Week 16 was chosen for the primary endpoint evaluations, as it will allow enough time for deucravacitinib to treat psoriasis and is the endpoint used in preceding psoriasis Phase 3 studies. The purpose of doing a 52-week study is to demonstrate the maintenance of improvement in PROs and clinical response.

A randomized, double-blind, placebo-controlled study provides the most robust assessment of efficacy and safety.



#### 6 STUDY POPULATION

Eligibility criteria for this study have been carefully considered to ensure: 1) selection of appropriate participants with psoriasis and 2) safety of the study participants. It is imperative that participants fully meet all eligibility criteria.

All screening and randomization evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

Prospective approval of protocol deviations to recruitment and enrollment criteria, also known as protocol waivers or exemptions, is not permitted.

#### 6.1 Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

#### 1) Signed Written Informed Consent

Participants must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written ICF in accordance with regulatory, local, and institutional guidelines. This must be obtained before the performance of any protocol-related procedures that are not part of normal patient care.

#### 2) Type of Participant and Target Disease Characteristics

- a) Men and women diagnosed with stable plaque psoriasis for 6 months or more. Stable psoriasis is defined as no morphology changes or significant flares of disease activity in the opinion of the investigator.
- b) Deemed by the investigator to be a candidate for phototherapy or systemic therapy
- c)  $\geq 3\%$  of BSA involvement at the Screening Visit and Day 1
- d) DLQI score > 5 at the Screening Visit and Day 1
- e) Moderate-to-severe plaque psoriasis Day 1

#### 3) Age of Participant

Participant must be  $\geq 18$  years of age inclusive at the time of signing the informed consent.

#### 4) Reproductive Status

Investigators shall counsel women of childbearing potential (WOCBP; as defined in APPENDIX 4) participants, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy.

The investigator shall evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

Local laws and regulations may require the use of alternative and/or additional contraception methods.

#### a) Female Participants:

- i) Women who are not of childbearing potential (as defined in APPENDIX 4) are exempt from contraceptive requirements.
- ii) WOCBP must have a negative highly sensitive serum pregnancy test at Screening Visit and a negative highly sensitive urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study intervention.
  - If a urine test cannot be confirmed as negative (eg, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
  - Additional requirements for pregnancy testing during and after study intervention are located in the Schedule of Activities (Section 2).
  - The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
- iii) WOCBP must agree to follow instructions for method(s) of contraception defined in APPENDIX 4 and as described below and included in the ICF.
- iv) WOCBP are permitted to use hormonal contraception methods (as described in APPENDIX 4)
- v) A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies:
  - (1) Is not a WOCBP OR
  - (2) Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with low user dependency, as described in APPENDIX 4, during the study period until the end of the study.

#### b) Male Participants:

i) Male participants should maintain their usual practice with regard to contraception (if any); however, no specific contraceptive measures are required.

#### 6.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

#### 1) Target Disease Exceptions

a) Has non-plaque psoriasis (ie, guttate, pustular, erythrodermic, palmoplantar only involvement or drug-induced psoriasis) at screening or Day 1

#### 2) Reproductive Status

- a) Women who are pregnant
- b) Women who are breastfeeding
- c) Women who are lactating
- d) Women who are planning pregnancy during the study period

#### 3) Infectious/Immune-related Exclusions

- a) History or evidence of outpatient active infection and/or febrile illness within 7 days prior to Day 1
- b) History of serious bacterial, fungal, or viral infection requiring hospitalization and/or intravenous antimicrobial intervention within 60 days prior to Day 1
- c) Any untreated bacterial infection within 60 days prior to Day 1
- d) Any ongoing evidence of chronic, bacterial infection (eg, chronic pyelonephritis, chronic osteomyelitis, chronic bronchiectasis)
- e) Any history of proven infection of a joint prosthesis in which the prosthesis was not removed or replaced, or received antibiotics for suspected infection of a joint prosthesis in which the prosthesis was not removed or replaced
- f) Not applicable per Protocol Amendment 02: Participants who are not fully vaccinated against SARS-CoV-2 as defined by the local and current national guidelines
- g) Received live vaccines within 60 days prior to Day 1, or plans to receive a live vaccine during the study, or within 60 days after completing study intervention
- h) Receipt of any non-live vaccine within 30 days prior to Day 1 including any COVID-19 vaccine (first, second or booster dose)
- i) Presence of herpes zoster lesions at screening or Day 1
- j) History of serious herpes zoster or serious herpes simplex infection which includes, but is not limited to, any episode of disseminated herpes simplex, multi-dermatomal herpes zoster, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (recurrent is defined as 2 episodes within 2 years)
- k) Evidence of, or test positive for, hepatitis B virus at Screening. Positive hepatitis B lab testing is defined as (please see APPENDIX 6 for details):
  - i) Positive hepatitis B surface antigen (HBsAg+)

#### OR

ii) Not applicable per Protocol Amendment 02: Presence of hepatitis B virus deoxyribonucleic acid (DNA)

#### OR

- 1) Evidence of, or test positive for, hepatitis C virus (HCV) at screening. A positive test for HCV is defined as: 1) positive for hepatitis C virus antibody AND 2) positive via a confirmatory test for HCV (eg, HCV polymerase chain reaction)
- m) Positive for human immunodeficiency virus (HIV) by antibody testing (HIV-1 and HIV-2 antibody) at screening
- n) Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status (eg, history of opportunistic infections [eg, *Pneumocystis jirovecii* pneumonia, histoplasmosis, or coccidioidomycosis], history of splenectomy, primary immunodeficiency)
- o) Severe SARS-CoV-2 infection within 4 weeks prior to screening. Additionally, in the case of prior SARS-CoV-2 infection, symptoms must have completely resolved and based on investigator assessment in consultation with the clinical study physician, there are no sequelae that would place the participant at a higher risk of receiving investigational intervention.

#### 4) Any of the following TB criteria

- a) Participant has a history of active TB prior to Screening Visit, regardless of completion of adequate treatment
- b) Participant has signs or symptoms of active TB (eg, fever, cough, night sweats, and weight loss) during Screening as judged by the investigator





#### 5) Medical History and Concurrent Diseases

- a) Any major surgery within 8 weeks prior to Day 1, or any planned major surgery for the first 52 weeks of the study
- b) Drug or alcohol abuse, as determined by the investigator, within 6 months prior to Day 1
- c) Medical marijuana or prescription marijuana taken for medicinal reasons
- d) Any major illness/condition or evidence of an unstable clinical condition (eg, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, psychiatric, neurologic, immunologic, or local active infection/infectious illness) that, in the investigator's judgement or after consultation with the Medical Monitor or designee, will substantially increase the risk to the participant if he or she participates in the study
- e) Unstable cardiovascular disease, defined as a recent clinical cardiovascular event (eg, unstable angina, myocardial infarction, stroke, rapid atrial fibrillation) in the last 3 months prior to screening, or a cardiac hospitalization (eg, revascularization procedure, pacemaker implantation) within 3 months prior to screening
- f) Has uncontrolled arterial hypertension characterized by a systolic blood pressure (BP) > 160 mm Hg or diastolic BP > 100 mm Hg
  - Note: Determined by 2 consecutive elevated readings. If an initial BP reading exceeds this limit, the BP may be repeated once after the participant has rested sitting for  $\geq 10$  minutes. If the repeat value is less than the criterion limits, the second value may be accepted
- g) Class III or IV congestive heart failure by New York Heart Association criteria
- h) Has cancer or history of cancer (solid organ or hematologic including myelodysplastic syndrome) or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell or squamous cell carcinoma, or carcinoma of cervix in situ that has been treated with no evidence of recurrence)



- k) If the participant has received biologics previously, the following exclusion criteria for washout will apply:
  - i) Antibodies to IL-12, IL-17, or IL-23 (eg, ustekinumab, secukinumab, tildrakizumab, ixekizumab, or guselkumab, tildrakizumab and risankizumab) within 6 months of Day 1
  - ii) TNF inhibitor(s) (eg, etanercept, adalimumab, infliximab, certolizumab) within 2 months of Day 1
  - iii) Agents that modulate integrin pathways to impact lymphocyte trafficking (eg, natalizumab), or agents that modulate B cells or T cells (eg, alemtuzumab, abatacept, or visilizumab) within 3 months of Day 1
  - iv) Rituximab within 6 months of Day 1
- 1) Has received systemic non-biologic psoriasis medications and/or any systemic immunosuppressants (including, but not limited to, methotrexate, azathioprine, cyclosporine, JAK inhibitors, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus, oral or injectable corticosteroids, retinoids, psoralens, sulfasalazine, or fumaric acid derivatives and apremilast) within 4 weeks prior to Day 1
- m) Has used leflunomide within 6 months prior to Day 1
- n) Has used opioid analgesics within 4 weeks prior to Day 1
- o) Has received lithium, antimalarials, or intramuscular gold within 4 weeks of the first administration of any study medication
- p) Has received phototherapy (including either oral and topical psoralens with ultraviolet A light therapy, ultraviolet B, or self-intervention with tanning beds or therapeutic sunbathing) within 4 weeks prior to Day 1
- q) Has used topical medications/interventions that could affect psoriasis evaluation (including, but not limited to, high potency corticosteroids [World Health Organization (WHO) Classes I to V], > 3% salicylic acid, urea, alpha- or beta-hydroxyl acids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, pimecrolimus, and tacrolimus) and intralesional corticosteroids within 2 weeks prior to Day 1
- r) Use of shampoos that contain corticosteroids, coal tar, > 3% salicylic acid, or vitamin D<sub>3</sub> analogues within 2 weeks prior to Day 1
- s) Has received an experimental antibody or experimental biologic therapy within the previous 6 months, OR received any other experimental therapy or new investigational agent, including those for SARS-CoV-2, within 30 days or 5 half-lives (whichever is longer) prior to Day 1 OR is currently enrolled in an investigational study

t) Any other sound medical, psychiatric and/or social reasons as determined by the investigator

## 6) Physical and Laboratory Test Findings

- a) At Screening
  - i) Absolute white blood cell count < 3000/mm<sup>3</sup>
  - ii) Absolute lymphocyte count < 500/mm<sup>3</sup>
  - iii) Absolute neutrophil count < 1000/mm<sup>3</sup>
  - iv) Platelet count < 100,000/mm<sup>3</sup>
  - v) Hemoglobin < 9 g/dL
  - vi) Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN)
  - vii) Total, unconjugated, and/or conjugated bilirubin > 2 × ULN
- b) Electrocardiograms (ECG) abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if participating in the study
- c) Inability to be venipunctured and/or tolerate venous access
- d) Any other significant laboratory abnormalities that, in the opinion of the investigator, might place the participant at unacceptable risk for participation in this study

#### 7) Allergies and Adverse Drug Reaction

a) History of any significant drug allergy (such as anaphylaxis)

#### 8) Other Exclusion Criteria

- a) Prisoners or participants who are involuntarily incarcerated. (Note: Under certain specific circumstances and only in countries where local regulations permit, a person who has been imprisoned may be included or permitted to continue as a participant. Strict conditions apply, and BMS approval is required)
- b) Participants who are compulsorily detained for intervention of either a psychiatric or physical (eg, infectious disease) illness
- c) Inability to comply with restrictions and prohibited activities/interventions as listed in the study protocol
- d) Participation in another clinical study concurrent with this study

Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

#### 6.3 Lifestyle Restrictions

General skin care measures (with above restrictions for topical interventions) are recommended that are standard for participants with plaque psoriasis. Participants should avoid excessive sun exposure or use of tanning booths or other UV light sources and avoid risks that are known to provoke flare of psoriasis.

#### 6.3.1 Meals and Dietary Restrictions

Study intervention may be taken without regard to meals;

#### 6.3.2 Caffeine, Alcohol and Tobacco

No restrictions are required; however, extensive use of caffeine, alcohol, tobacco, and vaping should be avoided.

#### 6.3.3 Activity

No restrictions are required.

#### 6.4 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but who are not subsequently randomized in the study/included in the analysis population.

A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants, to meet the Consolidated Standards of Reporting Trials publishing requirements, as applicable, and to respond to queries from regulatory authorities. Minimal information includes date of consent, demography, screen failure details, eligibility criteria, and any serious AEs.

## 6.4.1 Retesting During the Screening Period

For laboratory parameters that initially do not meet eligibility requirements, a single retest within the 28-day screening period is permitted before participant is declared a screen failure. This is an effort to find all possible well-qualified participants. Consultation with the Medical Monitor or designee may be needed to identify whether repeat testing of any parameter would be clinically relevant.

The study permits the rescreening (after the end of the initial 28-day screening period) of a participant who discontinues the study as a pretreatment failure (ie, the participant fails to meet eligibility criteria and has not been treated). If re-enrolled, the participant must be reconsented, assigned a new identification number, and a full Screening Visit must be performed again. A participant can only be rescreened 1 time (ie, if the participant fails 1 rescreening attempt, no additional rescreening is allowed). Depending on the timing of rescreening, repetition of some assessments may not be required. The fewest number of procedures from the initial screening should be repeated to qualify the participant, while maintaining participant safety and eligibility. In these cases, the site should consult with the BMS Medical Monitor (or designee).

Duration of existing interventions and required discontinuation periods shall be considered relative to the new Screening Visit and/or randomization.

The most current result(s) prior to randomization is the value by which study inclusion will be assessed, because it represents the participant's most current clinical state.

#### 7 STUDY INTERVENTION(S) AND CONCOMITANT THERAPY

Study intervention is defined as any investigational intervention(s), marketed product(s), placebo, procedure(s) or medical device intended to be administered to a study participant according to the study protocol.

Study intervention includes both investigational [medicinal] product (IP/IMP) and non-investigational [medicinal] product (non-IP/non-IMP) as indicated in Table 7.1-1.

An IP, also known as IMP in some regions, is defined as a pharmaceutical form of an active substance or placebo being tested or used as a reference in a clinical study, including products already with a marketing authorization but used or assembled (formulated or packaged) differently from the authorized form, or used for an unauthorized indication, or when used to gain further information about the authorized form.

Other medications used as support or escape medication for preventative, diagnostic, or therapeutic reasons, as components of the standard of care for a given diagnosis, may be considered as non-IPs.

# 7.1 Study Interventions Administered

The selection and timing of dose for each participant is presented in in Table 7.1-1.

**Table 7.1-1:** Study Interventions

| Arm Name | Deucravacitinib<br>(BMS-986165) | Placebo |
|---|---|---|
| Intervention Name | Deucravacitinib (BMS-986165) | Placebo for deucravacitinib |
| Туре | Drug | Drug |
| Dose Formulation | Tablet | Placebo tablet to match deucravacitinib |
| Unit Dose Strength(s) | 6 mg | n/a |
| Dosage Level(s) | 1 active tablet QD in the morning | 1 placebo QD in the morning |
| Route of Administration | Oral | Oral |
| Use | Experimental | Placebo |
| IMP and NIMP/AxMP | IMP | IMP |
| Sourcing | Provided centrally by the Sponsor | Provided centrally by the Sponsor |
| Packaging and Labeling | Study intervention will be provided in a bottle. Each bottle will be labeled as required per country requirement. | Study intervention will be provided in a bottle. Each bottle will be labeled as per country requirement. |

AxMP, auxiliary medicinal products; IMP, investigational medicinal product; n/a, not applicable; NIMP, non-investigational medicinal product; QD, once daily.

## 7.2 Method of Study Intervention Assignment

Before the study is initiated, each user (at investigative sites) will receive log-in information and directions on how to access the IRT system. At the time of the Screening Visit, immediately after informed consent is obtained and before any study-related procedures are performed, the investigative site will access the enrollment option of the IRT system for assignment of a participant number for all participants, including participants not subsequently randomized or treated. The participant number is assigned sequentially by the system and will be unique across all sites. All enrolled participants will be assigned sequential participant numbers. The participant number will not be used for any other participant. If a participant is rescreened, they will be given a new identification number.

At Day 1, participants who meet all criteria for enrollment at Screening and Day 1 will be centrally randomized in a 2:1 ratio to deucravacitinib 6 mg QD or placebo as determined by a computer-generated randomization schedule using IRT. The randomization lists will be generated by the IRT vendor using a permuted block design within each stratum level.

After all inclusion/exclusion criteria have been met for a participant, the investigative site will access the IRT on Day 1 for the purpose of randomizing a participant. An intervention group will be assigned by IRT based on the above-described randomization schedule. In addition, a unique kit number will be assigned to the participant corresponding to the intervention assignment.

Study intervention will be dispensed at study visits as shown in the Schedule of Activities (Section 2). When new intervention kits need to be provided, the investigative site will access the IRT to obtain the kit number to assign to the participant.

At Week 16, all participants, regardless of their blinded intervention, will be switched to open-label deucravacitinib 6 mg QD bottles through Week 52.

#### 7.3 Blinding

This is a randomized, double-blind, placebo-controlled study.

#### 7.3.1 Maintaining the Blind

Blinded intervention assignments will be managed using IRT. IP supply will be controlled by IRT at each visit.

All tablets are identical in appearance and will be supplied in bottles with each daily dose made up of the appropriate combination of active and/or placebo tablets to provide the correct intervention, as shown in Table 7.1-1. Investigative site staff, Sponsor and designee personnel, and participants and their families will remain blinded to intervention assignments.

The Sponsor and site facing study team will be unblinded to the individual treatment assignments at the primary endpoint database lock after the last participant has completed the Week 16 visit.

Clinical Protocol BMS-986165

The primary analysis database lock will occur after all randomized participants completed their Week 16 visit or discontinued prior to Week 16. The study participants and investigators will remain blinded to the initial treatment assignment throughout the study.

## 7.3.2 Circumstances for Unblinding

Blinding of study treatment assignment is critical to the integrity of this clinical study. However, in the event of a medical emergency or pregnancy in an individual participant in which knowledge of the IP is critical to the participant's management, the blind for that participant may be broken by the investigator. The participant's safety takes priority over any other considerations in determining if a treatment assignment should be unblinded.

Before breaking the blind of an individual participant's treatment, the investigator should determine that the unblinded information is necessary (ie, that it will alter the participant's immediate management). In many cases, particularly when the emergency is clearly not related to the IP, the problem may be properly managed by assuming that the participant is receiving the IP.

It is highly desirable that the decision to unblind treatment assignment be discussed with the Medical Monitor, but the investigator always has ultimate authority for the decision to unblind. The actual task of unblinding can be delegated by the investigator to a designee assigned the task on the Delegation of Authority. The Principal Investigator or appointed designee should only call in for emergency unblinding after the decision to unblind the participant has been documented.

For this study, the method of unblinding for emergency purposes is described in the IRT manual.

In case of an emergency, the investigator has unrestricted access to randomization information via IRT and is capable of breaking the blind through the IRT system without prior approval from the Sponsor. After the unblinding, the investigator shall notify the Medical Monitor or designee and/or study director. Participant and unblinded treatment information and the reason for the blind being broken must be recorded on the appropriate study status page of the eCRF. After unblinding via IRT, the investigator shall notify the Medical Monitor or designee.

In cases of accidental unblinding, contact the Medical Monitor and ensure every attempt is made to minimize additional disclosure and the impact of unblinding.

Any request to unblind a participant for nonemergency purposes should be discussed with the Medical Monitor.

If a participant is unblinded for any reason, the participant will be discontinued from treatment.

## 7.4 Dosage Modification

There is no provision for dose modification of study intervention. If a participant interrupts intervention due to an AE, study intervention can be restarted in consultation with the Medical Monitor or designee.

# 7.5 Preparation/Handling/Storage/Accountability

The IP must be stored in a secure area according to local regulations. It is the responsibility of the investigator, or designee where permitted, to ensure that IP is only dispensed to study participants.

Clinical Protocol BMS-986165 IM011237 Deucravacitinib

The IP must be dispensed only from official study sites by authorized personnel according to local regulations.

The product storage manager should ensure that the study intervention is stored in accordance with the environmental conditions (temperature, light, and humidity) as determined by BMS. If concerns regarding the quality or appearance of the study intervention arise, the study intervention should not be dispensed, and BMS should be contacted immediately.

Study intervention not supplied by BMS will be stored in accordance with the package insert.

IP documentation (whether supplied by BMS or not) must be maintained that includes all processes required to ensure the drug is accurately administered. This includes documentation of drug storage, administration and, as applicable, storage temperatures, reconstitution, and use of required processes (eg, required diluents, administration sets).

- The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study intervention received and any discrepancies are reported and resolved before use of the study intervention.
- The investigator, institution, or the head of the medical institution (where applicable) is responsible for study intervention accountability, reconciliation, and record maintenance (ie, receipt, reconciliation, and final disposition records).
- Further guidance and information for the final disposition of unused study interventions are provided in the Study Reference Manual.

#### 7.6 Treatment Compliance

When participants self-administer study intervention(s) at home, compliance with study intervention will be assessed at each visit. Compliance will be assessed by direct questioning, counting returned tablets, etc, during the site visits and documented in the source documents and relevant form. Deviation(s) from the prescribed dosage regimen should be recorded in the Case Report Form (CRF).

A record of the quantity of deucravacitinib/placebo dispensed to and administered by each participant must be maintained and reconciled with study intervention and compliance records. Intervention start and stop dates, including dates for intervention delays and/or dose reductions, will also be recorded in the CRF.

# 7.7 Concomitant Therapy

#### 7.7.1 Prohibited and/or Restricted Treatments

Prohibited and/or restricted medications taken during the study are described below.

- Exposure to any investigational drug, investigational vaccine, or placebo outside of the current study. Specifically, participants currently in other interventional studies for COVID-19, including investigational COVID-19 vaccination studies that are not authorized or approved by relevant Health Authorities, should not participate in BMS clinical studies
- Use of any medications/therapy that would aggravate psoriasis. These include agents such as lithium, antimalarials (quinacrine, chloroquine, and hydroxychloroquine), propranolol,

indomethacin, and quinidine unless it is considered necessary for the participant's welfare and/or intervention of an AE/SAE

- Use of opioid analgesics unless it is considered necessary for the participant's welfare and/or treatment of an AE/SAE
- Phototherapy; use of tanning booths or therapeutic sunbathing
- Any use of biologic medications (eg, adalimumab, etanercept, infliximab, ustekinumab).
- Any use of oral psoriasis medications (eg, apremilast, methotrexate, cyclosporine, retinoids, fumaric acid derivatives) for any indication
- Any use of oral or injectable corticosteroids (prednisone, methylprednisolone, etc), unless it is
  considered necessary for the participant's welfare and/or intervention of an AE/SAE
  Note: optic, ophthalmic, nasal, and inhaled corticosteroids within recommended doses and
  with no systemic effects are permitted.
- Any topical medications/interventions, which are used for any indication, that could affect psoriasis evaluation (including, but not limited to, high potency corticosteroids [WHO Classes I to V], > 3% salicylic acid, urea, alpha- or beta-hydroxy acids, anthralin, calcipotriene, vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, pimecrolimus, and tacrolimus) and intralesional corticosteroids.



- Any medicated shampoos that contain corticosteroids, coal tar, > 3% salicylic acid, or vitamin D<sub>3</sub> analogues
- Live attenuated vaccines (including, but not limited to, any live attenuated COVID-19 vaccines) should not be used during the study, including the safety follow-up period of 60 days following last dose of IP (see Section 7.7.4 for permitted vaccines).

#### 7.7.2 Permitted Concomitant Medications

Participants may take any medication that is not restricted by the protocol, is not expected to interfere with the conduct of the study and will not affect study assessments. Stable doses of concomitant medication for chronic medical conditions are permitted if neither the medication nor the medical condition meet exclusion criteria as detailed in Section 6.2. Dose adjustments of these

medications should be avoided during the study unless clinically indicated. If a dose adjustment of these medications should occur, they must be recorded on the Concomitant Medications eCRF. The investigator should instruct the participant to notify the study site about any new treatment he/she takes after the start of the study intervention. All medications and significant nondrug therapies (including physical therapy and blood transfusions) administered after the participant starts study intervention must be listed on the Concomitant Medications eCRF.

Concomitant medications (prescription, over the counter, or herbal) should be administered during the study only if they are to be used for treatment of specific medical reasons.



# 7.7.4 Permitted Vaccines (Including COVID-19 Vaccine)

Administration of a non-live vaccine is allowed during the study. However, the efficacy and safety of non-live vaccines (including non-live COVID-19 vaccines) in participants receiving deucravacitinib is unknown. The following are examples of non-live vaccines: inactivated vaccines (eg, heat-killed and formalin-killed vaccines), subunit vaccines (eg, influenza and pneumococcal vaccines), toxoid vaccines, nucleic acid vaccines that do not encode potentially infectious virus (eg, Pfizer/BioNTech and Moderna COVID-19 vaccines) and replication-incompetent recombinant vector vaccines (eg, AstraZeneca/University of Oxford COVID-19 vaccine).

For COVID-19 vaccines requiring more than 1 dose, the full series (eg, both doses of a 2-dose series) should be completed 30 days prior to enrollment. Ideally, AEs attributable to a vaccine should have resolved prior to enrollment.

If a participant receives a COVID-19 vaccination during the study, details such as type and date of vaccine received should be recorded on the concomitant medication page. For COVID-19 vaccines administered prior to enrollment, the types, details, and dates should be also recorded on the appropriate eCRF page.

Please contact the Medical Monitor or designee with any questions related to COVID-19 vaccines.

#### 7.8 Continued Access to Study Intervention After the End of the Study

At the end of the study, BMS will not continue to provide BMS-supplied study intervention to participants/investigators unless BMS chooses to extend the study. The investigator should ensure that participant receives appropriate standard of care to treat the condition under study.

#### 8 DISCONTINUATION CRITERIA

## 8.1 Discontinuation From Study Intervention

Participants MUST discontinue IP/IMP for any of the following reasons:

- Participant's request to stop study intervention. Participants who request to discontinue study intervention will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him/her or persons previously authorized by the participant to provide this information
- Any clinical AE, laboratory abnormality, or intercurrent illness which, in the opinion of the investigator, indicates that continued participation in the study is not in the best interest of the participant
- Termination of the study by BMS
- Loss of ability to freely provide consent through imprisonment or involuntarily incarceration for treatment of either a psychiatric or physical (eg, infectious disease) illness.
  - Note: Under specific circumstances and only in countries where local regulations permit, a participant who has been imprisoned may be permitted to continue as a participant. Strict conditions apply, and BMS approval is required
- Abnormal liver tests suggestive of drug-induced liver injury (DILI), as defined in Section 9.2.8 or if the investigator believes that it is in the best interest of the participant
- The participant develops a malignancy, with the exception of a participant who develops non-melanoma skin cancer who may continue in the study at the discretion of the investigator
- Pregnancy, positive pregnancy test or participant expresses an interest in becoming pregnant (Section 9.2.6)
- Unblinding of a participant's intervention assignment for any reason (emergency or nonemergency)
- Inability or failure to comply with protocol requirements in the opinion of the investigator
- Participant reports suicidal ideation, suicidal behavior, or suicide attempts at any time after inclusion. The participant should then be immediately referred to a mental health professional for evaluation of suicide risk

Refer to the Schedule of Activities (Section 2) for data to be collected at the time of intervention discontinuation and follow-up and for any further evaluations that can be completed.

In the case of pregnancy, the investigator must immediately, within 24 hours of awareness of the pregnancy, notify the BMS Medical Monitor/designee of this event. The study treatment will be permanently discontinued. See Section 8.

All participants who discontinue study intervention should comply with protocol-specified follow-up procedures as outlined in Section 2. The only exception to this requirement is when a participant withdraws consent for all study procedures, including post-treatment study follow-up, or loses the ability to consent freely (eg, is imprisoned or involuntarily incarcerated for the intervention of either a psychiatric or physical illness).

If study intervention is discontinued prior to the participant's completion of the study, the reason for the discontinuation must be documented in the participant's medical records per local regulatory requirements in each region/country and entered on the appropriate CRF page.

#### 8.1.1 Temporary Discontinuation from Study Intervention

Temporary study intervention discontinuation is only allowed if the participant develops an AE which, in the opinion of the investigator, indicates that it is in the participant's best interest that the study intervention be placed on hold. Study intervention in this situation should be stopped until the AE is medically treated and has resolved per investigator's judgement.

Temporary interruption of study treatment should be implemented in the context of clinical suspicion for SARS-CoV-2 or a positive diagnostic test for SARS-CoV-2. When study treatment is interrupted in a confirmed case of SARS-CoV-2, the investigator, in consultation with the Medical Monitor, should determine whether the resolution of symptoms alone (ie, without repeat diagnostic testing for SARS-CoV-2) is sufficient to resume study treatment.

Temporary interruption of study intervention may be considered in the event of SARS-CoV-2 vaccination according to local guidelines. To facilitate reporting of SARS-CoV-2 events that occur during the study, all AEs and SAEs related to SARS-CoV-2 must be reported from the time of consent. In addition, AEs or SAEs will trigger additional data collection through dedicated eCRF pages, which will allow the Sponsor to further evaluate these events.

Any temporary study intervention discontinuation as well as restart must be documented on the corresponding eCRF.

## 8.1.2 Post-Study Intervention Study Follow-up

In this study, efficacy is a key endpoint of the study. Post-study follow-up is of critical importance and is essential to preserving participant safety and the integrity of the study. Participants who discontinue study intervention must continue to be followed in this study for collection of outcome data as required and in line with Section 5 until the conclusion of the study.

## 8.2 Discontinuation From the Study

Participants who request to discontinue study intervention will remain in the study and must continue to be followed for protocol-specified follow-up procedures. The only exception to this is when a participant specifically withdraws consent for any further contact with him/her or persons previously authorized by participant to provide this information.

- Participants should notify the investigator of the decision to withdraw consent from future follow-up.
- The withdrawal of consent should be explained in detail in the medical records by the investigator, as to whether the withdrawal is from further treatment with study intervention only or also from study procedures and/or post-treatment study follow-up, and entered on the appropriate CRF page.
- In the event that vital status (whether the participant is alive or dead) is being measured, publicly available information should be used to determine vital status only as appropriately directed in accordance with local law.
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

#### 8.2.1 Individual Discontinuation Criteria

- A participant may withdraw completely from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons. This is expected to be uncommon. Stopping study intervention is not considered withdrawal from the study.
- At the time of discontinuing from the study, if possible, an early termination visit should be conducted, as shown in the Schedule of Activities (Section 2). See the Schedule of Activities (Section 2) for data to be collected at the time of study discontinuation and follow-up and for any further evaluations that need to be completed.
- The participant will be permanently discontinued both from the study intervention and from the study at that time.
- If the participant withdraws consent for disclosure of future information, the Sponsor may retain and continue to use any data collected before such a withdrawal of consent.

#### 8.3 Lost to Follow-up

The following actions must be taken if a participant fails to return to the clinic for a required study visit:

- All reasonable efforts must be made to locate participants to determine and report their ongoing status. This includes follow-up with persons authorized by the participant.
- Lost to follow-up is defined by the inability to reach the participant after a minimum of **3** documented phone calls, faxes, or emails, as well as lack of response by participant to 1 registered mail letter. All attempts should be documented in the participant's medical records.
- If it is determined that the participant has died, the site will use permissible local methods to obtain date and cause of death.
- If the investigator's use of third-party representative to assist in the follow-up portion of the study has been included in the participant's informed consent, then the investigator may use a Sponsor-retained third-party representative to assist site staff with obtaining the participant's contact information or other public vital status data necessary to complete the follow-up portion of the study.

Clinical Protocol BMS-986165 Deucravacitinib

The site staff and representative will consult publicly available sources, such as public health registries and databases, in order to obtain updated contact information.

• If, after all attempts, the participant remains lost to follow-up, then the last known alive date as determined by the investigator should be reported and documented in the participant's medical records.

#### 9 STUDY ASSESSMENTS AND PROCEDURES

- Study procedures and timing are summarized in the Schedule of Activities (Section 2).
- Protocol waivers or exemptions are not allowed.
- All immediate safety concerns must be discussed with the Sponsor immediately upon occurrence or awareness to determine if the participant should continue or discontinue intervention.
- Adherence to the study design requirements, including those specified in the Schedule of Activities (Section 2), is essential and required for study conduct.
- All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria before randomization. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.
- Procedures conducted as part of the participant's routine clinical management (eg, blood count) and obtained before signing of informed consent may be utilized for screening or baseline purposes provided the procedure meets the protocol-defined criteria and has been performed within the timeframe defined in the Schedule of Activities (Section 2).
- For several assessments, appropriate training will be provided to investigators and designated personnel at sites. Only those individuals trained and certified to perform these assessments will be performing them during the study.
- Repeat or unscheduled samples may be taken for safety reasons or for technical issues with the samples.

#### 9.1 **Efficacy Assessments**

Every effort must be made to ensure that the same evaluator(s) complete the assessment for each participant. If the evaluator(s) is/are unable to complete the evaluation, then a qualified individual with overlapping experience may perform the evaluation. Documentation of who performed the evaluation is to be recorded in source documents. Assessments are to be performed at approximately the same time of day throughout the duration of the study.

Baseline assessments must be performed per protocol (standard of care assessments may not be used for baseline). Procedures not specified in the protocol that are part of standard care may be performed if they do not interfere with study procedures; any data arising from such procedures are not to be reported in the eCRF.

Protocol Amendment 02 Date: 25-May-2023

IM011237

## 9.1.1 Investigator-Administered Assessments

#### 9.1.1.1 Static Physician's Global Assessment (s-PGA)

The s-PGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration.<sup>27</sup> The s-PGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). All s-PGA assessments should be performed by a trained physician (eg, dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients. Every effort should be made to ensure that the physician or designee who performed the s-PGA evaluations for a participant at randomization performs the s-PGA for that participant at all subsequent visits.

#### 9.1.1.2 Psoriasis Area and Severity Index (PASI)

The PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0–4 scale), weighted by the area of involvement (head, arms, trunk to groin, and legs to top of buttocks). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. The PASI can also be used to assess response to treatment. The PASI 50 is the proportion of participants who experience at least a 50% improvement in PASI score as compared with the baseline value. The PASI 75, PASI 90, and PASI 100 are defined similarly. BMS will host a training session prior to initiation of the study to demonstrate proper PASI scoring. All PASI assessments should be performed by a trained physician (dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients.

# 9.1.1.3 Body Surface Area (BSA)

Measurement of psoriasis BSA involvement is estimated using the handprint method with the size of a participant's handprint (including fingers and thumb) representing 1% of BSA involved. <sup>29,30,31</sup> The total BSA = 100% with breakdown by body region as follows:

Head and neck = 10% (10 handprints), upper extremities = 20% (20 handprints), trunk including axillae and groin = 30% (30 handprints), lower extremities including buttocks = 40% (40 handprints).

All BSA assessments should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients.

## 9.1.1.4 Scalp-Specific Physician's Global Assessment (ss-PGA)

For this assessment in participants with scalp involvement,<sup>32</sup> scalp lesions are evaluated in terms of clinical signs of redness, thickness, and scaliness and scored on the following 5-point ss-PGA scale:

```
0 = absence of disease, 1 = very mild disease, 2 = mild disease, 3 = moderate disease, 4 = severe disease.
```

The ss-PGA should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients.

## 9.1.1.5 Physician Global Assessment-Fingernails (PGA-F)

In this assessment,<sup>33</sup> the overall condition of the fingernails is rated on a 5-point scale:

```
0 = \text{clear}, 1 = \text{minimal}, 2 = \text{mild}, 3 = \text{moderate}, and 4 = \text{severe}.
```

The Physician Global Assessment-Fingernails (PGA-F) will be performed only in participants with psoriatic fingernail involvement to assess severity and subsequent improvement. The PGA-F should be performed by a dermatologist or appropriately training investigator who is experienced in the assessment of psoriasis patients.

#### 9.1.1.6 Palmoplantar PGA (pp-PGA)

This measure will be used for participants with palmoplantar involvement.<sup>34</sup> The palmoplantar Physician Global Assessment (pp-PGA) uses a 5-point (0-4) scale:

```
0 = \text{clear}; 1 = \text{almost clear}; 2 = \text{mild}; 3 = \text{moderate}; and 4 = \text{severe}.
```

The pp-PGA should be performed by a dermatologist or appropriately trained investigator who is experienced in the assessment of psoriasis patients.

# 9.1.1.7 Intertriginous-area s-PGA (I-s-PGA)

The intertriginous-area s-PGA (I-s-PGA) is a 5-point scale of an average assessment of intertriginous psoriatic lesions based on erythema, scale, and induration.<sup>35</sup> It is not necessary that all 3 criteria be fulfilled. The I-s-PGA score is based on a combination of erythema and the secondary features (plaque elevation and/or scale). Since erythema is the most robust finding, it should be the dominant feature influencing the I-s-PGA rating in the majority of cases. This intertriginous-area specific s-PGA measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). Intertriginous skin, also known as skin folds, are sites in which opposing skin surfaces come into contact while at rest, resulting in chronic skin occlusion. The primary intertriginous skin areas include the groin folds, axillae, gluteal cleft and perianal area. Body habitus may contribute to additional intertriginous sites, such as inframammary skin and abdominal folds. All I-s-PGA assessments should be performed by a trained physician (eg, dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients. Every effort should be made to ensure that the physician or designee who

performed the I-s-PGA evaluations for a participant at randomization performs the I-s-PG for that participant at all subsequent visits.

#### 9.1.1.8 s-PGA of Genitalia (s-PGA-G)

The s-PGA of Genitalia (s-PGA-G) is the clinician's determination of the participant's psoriasis lesions' overall severity in the genital area (labia majora, labia minora, and perineum in females; penis, scrotum, and perineum in males) at a given timepoint. Overall, lesions are categorized by descriptions for elevation, erythema, and scaling.<sup>36</sup> It is not necessary that all 3 criteria be fulfilled. The s-PGA-G score is based on a combination of erythema and the secondary features (plaque elevation and/or scale). Since erythema is the most robust finding, it should be the dominant feature influencing the s-PGA-G rating in the majority of cases. For the analysis of responses, the patient's psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). All s-PGA-G assessments should be performed by a trained physician (eg, dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients. Every effort should be made to ensure that the physician or designee who performed the s-PGA-G evaluations for a participant at randomization performs the s-PGA-G for that participant at all subsequent visits.

## 9.1.1.9 Static Physician Global Assessment for the Face (sf-PGA)

The static Physician Global Assessment for the face (sf-PGA) of face is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration only on the face. The sf-PGA of face measure determines psoriasis severity at a single point in time (without taking into account the baseline disease condition) as clear (0), almost clear (1), mild (2), moderate (3), or severe (4). All sf-PGA assessments should be performed by a trained physician (eg, dermatologist) or appropriately trained investigator who is experienced in the assessment of psoriasis patients. Every effort should be made to ensure that the physician or designee who performed the sf-PGA evaluations for a participant at randomization performs the sf-PGA for that participant at all subsequent visits.





Date: 25-May-2023





#### 9.2 Adverse Events

The definitions of an AE or SAE can be found in APPENDIX 3.

AEs will be reported by the participant (or, when appropriate, by a caregiver, or a surrogate, or the participant's legally acceptable representative). The investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up on AEs that are serious, considered related to the study intervention or the study, or that caused the participant to discontinue before completing the study.

Refer to APPENDIX 3 for SAE reporting.



## 9.2.2 Time Period and Frequency for Collecting AE and SAE Information

The collection of nonserious AE information should begin at initiation of study intervention until discharge from the study (ie, final study visit for a given participant), at the timepoints specified in the Schedule of Activities (Section 2).

Appendix 1 of the IB<sup>26</sup> represents the Reference Safety Information to determine expectedness of SAEs for expedited reporting.

All SAEs must be collected from the time of signing the consent, including those thought to be associated with protocol-specified procedures, and within 30 days following discontinuation of dosing.

The investigator must report any SAE that occurs after these time periods and that is believed to be related to study intervention or protocol-specified procedure.

- Medical occurrences that begin before the start of study intervention but after obtaining informed consent will be recorded on the appropriate section of the CRF module.
- All SAEs will be recorded and reported to Sponsor or designee within 24 hours, as indicated in APPENDIX 3.
- The investigator will submit any updated SAE data to the Sponsor or designee within 24 hours of updated information being available.

Investigators are not obligated to actively seek AEs or SAEs in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a participant has been discharged from the study, and he/she considers the event reasonably related to the study intervention or study participation, the investigator must promptly notify the Sponsor.

The method of evaluating and assessing causality of AEs and SAEs and the procedures for completing and reporting/transmitting SAE reports are provided in APPENDIX 3.

## 9.2.3 Method of Detecting AEs and SAEs

AEs can be spontaneously reported or elicited during open-ended questioning, examination, or evaluation of a participant. Care should be taken not to introduce bias when collecting AEs and/or SAEs. Inquiry about specific AEs should be guided by clinical judgement in the context of known AEs, when appropriate for the program or protocol.

# 9.2.4 Follow-up of AEs and SAEs

- Nonserious AEs should be followed to resolution or stabilization, or reported as SAEs if they become serious (see APPENDIX 3).
- Follow-up is also required for nonserious AEs that cause interruption or discontinuation of study intervention and for those present at the end of study intervention as appropriate.
- All identified nonserious AEs must be recorded and described on the nonserious AE page of the CRF (paper or electronic). Completion of supplemental CRFs may be requested for AEs and/or laboratory abnormalities that are reported/identified during the course of the study.

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs, will be

followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the participant is lost to follow-up (as defined in Section 8.3).

Further information on follow-up procedures is given in APPENDIX 3.

# 9.2.5 Regulatory Reporting Requirements for SAEs

- Prompt notification by the investigator to the Sponsor of SAEs is essential so that legal obligations and ethical responsibilities toward the safety of participants and the safety of a product under clinical investigation are met.
- An investigator who receives an investigator safety report describing SAEs or other specific safety information (eg, summary or listing of SAEs) from the Sponsor will file it along with the IB and will notify the IRB/IEC, if appropriate according to local requirements.

The Sponsor or designee must report AEs to regulatory authorities and ethics committees according to local applicable laws and regulations. A SUSAR (suspected, unexpected serious adverse reaction) is a subset of SAEs and must be reported to the appropriate regulatory authorities and investigators following local and global guidelines and requirements.

#### 9.2.6 Pregnancy

If, following initiation of the study intervention, it is subsequently discovered that a participant is pregnant or may have been pregnant at the time of study exposure, including during at least for 30 days after study product administration, the investigator must immediately notify the BMS Medical Monitor/designee of this event and complete and forward a Pregnancy Surveillance Form to the BMS designee within 24 hours of awareness of the event and in accordance with SAE reporting procedures described in APPENDIX 3.

Follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome and, where applicable, offspring information, must be reported on the Pregnancy Surveillance Form. Protocol-required procedures for study discontinuation and follow-up must be performed on the participant.

In the event a participant becomes pregnant during the study, the study intervention must be discontinued immediately.

#### 9.2.7 Laboratory Test Result Abnormalities

The following laboratory test result abnormalities should be captured on the nonserious AE CRF page or SAE eCRF, as appropriate. Paper forms are only intended as a back-up option when the electronic system is not functioning.

- Any laboratory test result that is clinically significant or meets the definition of an SAE
- Any laboratory test result abnormality that required the participant to have study intervention discontinued or interrupted
- Any laboratory test result abnormality that required the participant to receive specific corrective therapy

It is expected that, wherever possible, the clinical rather than laboratory term would be used by the reporting investigator (eg, anemia vs low hemoglobin value).

#### 9.2.8 Potential Drug-induced Liver Injury (DILI)

Wherever possible, timely confirmation of initial liver-related laboratory abnormalities should occur prior to the reporting of a potential DILI event. All occurrences of potential DILIs meeting the defined criteria must be reported as SAEs (see Section 9.2.5 and APPENDIX 3 for reporting details).

A potential DILI is defined as:

1) Aminotransferase (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) elevation > 3× ULN

#### **AND**

2) Total bilirubin > 2 × ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)

#### **AND**

3) No other immediately apparent possible causes of aminotransferase elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, pre-existing chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic.

## 9.2.9 Other Safety Considerations

Any significant worsening of conditions noted during interim or final PEs, ECG, x-ray filming, or any other potential safety assessment required or not required by the protocol should also be recorded as a nonserious AE or SAE, as appropriate, and reported accordingly.

#### 9.3 Overdose

For this study, any dose of deucravacitinib greater than 24 mg within a 24-hour time period will be considered an overdose. Overdoses that meet the regulatory definition of SAE will be reported as an SAE (see APPENDIX 3).

In the event of an overdose, the investigator should:

- 1) Contact the Medical Monitor or designee immediately
- 2) Closely monitor the participant for AEs/SAEs and laboratory abnormalities for at least 5 half-lives of deucravacitinib, approximately 3 days

Decisions regarding dose interruptions will be made by the investigator in consultation with the Medical Monitor or designee based on the clinical evaluation of the participant.

#### 9.4 Safety

Planned timepoints for all safety assessments are listed in the Schedule of Activities (Section 2).

## 9.4.1 Physical Examinations

A complete PE will include general appearance, vital signs, eyes, ears, nose, mouth, throat, neck, respiratory, cardiovascular, respiratory, gastrointestinal/abdomen, lymphatic, musculoskeletal, skin, psychiatric and neurologic exams. A targeted PE will include any organ system associated with an AE or a laboratory abnormality.
While the targeted PE may not be as comprehensive as the initial full examination, key aspects should evaluate important body systems as clinically indicated. These body systems can include lymph nodes, liver, spleen, and breast at the discretion of the examiner. A targeted examination may note any changes in the participant's condition (body systems) since the last assessment and does not preclude examination of any of the other body systems as clinically indicated. Every effort should be made to ensure the same evaluator will complete the examination for each participant at all visits throughout the study. Documentation of who performed the examination is to be recorded in source notes.

# 9.4.2 Vital Signs

Vital signs include (ear or oral) body temperature, respiratory rate, and seated BP and heart rate and will be recorded at each visit based on the Schedule of Activities (Section 2). BP and heart rate should be measured after the participant has been seated quietly for at least 5 minutes.

# 9.4.3 Electrocardiograms

A 12-lead ECG will be performed at the Screening Visit indicated in the Schedule of Activities (Section 2). The participant will remain supine for 5 to 10 minutes prior to the ECG and must have their lab work done after the tracing so that the ECG results remain as accurate as possible. The ECG results will be read by the primary study investigator or a designee.







Date: 25-May-2023



# 9.10 Health Economics OR Medical Resource Utilization and Health Economics

Health economics/medical resource utilization and health economics parameters will not be evaluated in this study.

#### 10 STATISTICAL CONSIDERATIONS

There are 2 population groups of interest in this study:

- Overall Population: All participants who were randomized to any treatment arm in the study.
- s-PGA  $\geq$  3 Sub-Population: All participants who were randomized to any treatment arm in the study s-PGA  $\geq$  3 at baseline.

The statistical hypotheses associated with the primary endpoint (DLQI 0/1) and the secondary endpoints (at least a 4-point reduction from baseline in DLQI, whole-body itch NRS score and s-PGA 0/1 [s-PGA  $\geq$  3 Sub-Population only]), will be formally tested in each population group

# 10.1 Statistical Hypotheses

The primary hypotheses for the study are that the odds of achieving DLQI 0/1 at Week 16 in participants receiving deucravacitinib 6 mg QD are improved compared to participants receiving placebo on both the Overall Population and s-PGA  $\geq$  3 Sub-Population.

The null hypotheses to be tested for the primary endpoint are the following:

- The odds of achieving DLQI 0/1 at Week 16 in participants receiving deucravacitinib 6 mg QD are the same as participants receiving placebo on the Overall Population.
- The odds of achieving DLQI 0/1 at Week 16 in participants receiving deucravacitinib 6 mg QD are the same as participants receiving placebo on the s-PGA ≥ 3 Sub-Population.

Key secondary endpoints and associated hypotheses will be tested in a hierarchical order only if both primary hypotheses achieved statistical significance. The null hypotheses corresponding to the key secondary endpoints are described below by population.

# Overall Population:

- The odds of achieving at least a 4-point reduction from baseline in DLQI at Week 16 in participants receiving deucravacitinib 6 mg QD are the same as participants receiving placebo.
- The mean change from baseline in whole-body itch NRS score at Week 16 in participants receiving deucravacitinib 6 mg QD is not different from participants receiving placebo.

# s-PGA ≥ 3 Sub-Population:

- The odds of achieving at least a 4-point reduction from baseline in DLQI at Week 16 in participants receiving deucravacitinib 6 mg QD are the same as participants receiving placebo.
- The mean change from baseline in whole-body itch NRS score at Week 16 in participants receiving deucravacitinib 6 mg QD is not different from participants receiving placebo.
- The odds of achieving s-PGA 0/1 with at least a 2-point reduction from baseline at Week 16 in participants receiving deucravacitinib 6 mg QD are the same as participants receiving placebo.









# 10.3 Analysis Sets

For purposes of analysis, the populations and analysis data sets are defined in Table 10.3-1.

Table 10.3-1: Populations and Analysis Data Sets

| Population | Description |
|---|---|
| Enrolled | All participants who sign informed consent. |
| Randomized (FAS) | All participants who were randomized to any treatment arm in the study. |
| Full Analysis Subgroup | All participants who were randomized to any treatment arm in the study and baseline s-PGA $\geq$ 3. |
| Safety | All randomized participants who take at least 1 dose of study intervention. Participants will be analyzed according to intervention received. |
| Defined Analysis Data Sets | Description |
| Analysis set for primary estimand of DLQI 0/1 | All randomized participants with baseline s-PGA $\geq$ 3; all available data up to Week 16 database lock. Participants who discontinue prior to Week 16 will be imputed as non-responders in the analysis dataset. Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| | All randomized participants; all available data up to Week 16 database lock. Participants who discontinue prior to Week 16 will be imputed as non-responders in the analysis dataset. Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| | All randomized participants with baseline s-PGA ≥ 3; all available data up to Week 16 database lock. Participants who discontinue prior to Week 16 will be imputed as non-responders in the analysis dataset. |

| Defined Analysis Data Sets | Description |
|---|---|
| Analysis set for secondary estimand of ≥ 4-point reduction in DLQI from baseline | Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| | All randomized participants; all available data up to Week 16 database lock. Participants who discontinue prior to Week 16 will be imputed as non-responders in the analysis dataset. Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| Analysis set for secondary estimand of whole-body itch NRS | All randomized participants; all available data up to Week 16 database lock. Participants who discontinue prior to Week 16 will be imputed using multiple imputation in the analysis dataset. Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| | All randomized participants with baseline s-PGA $\geq$ 3; all available data up to Week 16 database lock. Participants who discontinue prior to Week 16 will be imputed using multiple imputation in the analysis dataset. Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| Analysis set for secondary estimand of s-PGA 0/1 | All randomized participants with baseline s-PGA $\geq$ 3; all available data up to Week 16 database lock. Participants who discontinued prior to Week 16 will be imputed as non-responders in the analysis dataset. Following the intent-to-treat principle, participants will be analyzed according to the intervention group assigned at randomization. |
| Analysis set for safety | All safety events reported for all randomized participants who are exposed to study intervention. For participants who discontinue study intervention all post-discontinuation up to day 28 post last dose of study intervention will be included in the safety summaries. Participants will be analyzed according to intervention received. |

DLQI, Dermatology Life Quality Index; FAS, Full Analysis Set; NRS, Numerical Rating Scale; s-PGA, static Physician Global Assessment.

# 10.4 Statistical Analyses

The statistical analysis plan (SAP) will be developed and finalized before the primary analysis database lock and will describe the selection of participants to be included in the analyses, and procedures for accounting for missing, unused, and spurious data. Below is a summary of planned statistical analyses of the primary and secondary endpoints. A description of the participant population will be included in the clinical study report (CSR), including subgroups of age, gender, race and other study specific populations and demographic characteristics. A description of participant disposition will also be included in the CSR.

#### 10.4.1 General Considerations

Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified. Efficacy values will be summarized for all visits in which the variable is assessed. Baseline values are defined as the last non-missing value prior to the first dose of study drug unless otherwise indicated.

During the first 16 weeks of treatment, data will be presented for the following interventions:

- Deucravacitinib 6 mg QD
- Placebo

After Week 16, data will be presented for the following interventions:

- Deucravacitinib 6 mg QD
- Placebo- deucravacitinib 6 mg QD (starting at Week 16 through Week 52)

The primary endpoint, DLQI 0/1 response, is defined as a proportion of participants achieving DLQI score of 0 or 1 at Week 16. The key secondary endpoints assessed at Week 16 are  $\geq$  4-point reduction from baseline in DLQI, change from baseline in whole-body itch NRS score and s-PGA 0/1 response. s-PGA 0/1 is defined as a proportion of participants with a s-PGA score of 0 (clear) or 1 (almost clear) with at least a 2-point reduction from baseline at Week 16.

Table 10.4.1-1: Definition of Estimands for Primary and Key Secondary Endpoints

| Primary Endpoint | | | |
|---|---|---|---|
| Estimand Attribute | Definition | | |
| Treatment | Deucravacitinib 6 mg QD v | ersus placebo | |
| Population | FAS population and FAS su | b-population | |
| Variable | DLQI 0/1 | | |
| ICEs | Event | Strategy | Description |
| | Discontinuation of intervention or study early prior to Week 16 assessment | Composite variable | Participant will be counted as a non-responder |
| | Lost to follow-up prior to<br>Week 16 or otherwise<br>missing endpoint data at<br>Week 16 assessment | Composite variable | Participant will be counted as a non-responder |
| | Start a protocol prohibited medication/therapy | Treatment policy | Participants will be included in the primary analysis regardless of the occurrence of the ICE according to the respective endpoint definition. |
| | Missing assessment at<br>Week 16 due to<br>SARS-CoV-2 | While on treatment | Participants will be excluded from the primary analysis if the Week 16 assessment was not completed due to SARS-CoV-2 |
| Population-level<br>Summary | Odds ratio of achieving DLQI 0/1 | | |

Table 10.4.1-1: Definition of Estimands for Primary and Key Secondary Endpoints

| Key Secondary Endpoi | nts | | |
|---|---|---|---|
| <b>Estimand Attribute</b> | Definition | | |
| Treatment | Deucravacitinib 6 mg QD versus placebo | | |
| Population | FAS population and FAS su | ıb-population | |
| Variable | ≥ 4-point reduction from ba | seline in DLQI | |
| ICEs | Event | Strategy | Description |
| | Discontinuation of intervention or study early prior to Week 16 assessment | Composite variable | Participant will be counted as a non-responder |
| | Lost to follow-up prior to<br>Week 16 or otherwise<br>missing endpoint data at<br>Week 16 assessment | Composite variable | Participant will be counted as a non-responder |
| | Start a protocol prohibited medication/therapy | Treatment policy | Participants will be included in the analysis regardless of the occurrence of the ICE according to the respective endpoint definition. |
| | Missing assessment at<br>Week 16 due to<br>SARS-CoV-2 | While on treatment | Participants will be excluded from the analysis if the Week 16 assessment was not completed due to SARS-CoV-2 |
| Population-level<br>Summary | Odds ratio of achieving ≥ 4 | Odds ratio of achieving ≥ 4-point reduction from baseline in DLQI | |
| <b>Estimand Attribute</b> | Definition | | |
| Treatment | Deucravacitinib 6 mg QD v | ersus placebo | |
| Population | FAS population and FAS su | FAS population and FAS sub-population | |
| Variable | Change from baseline in wh | nole-body itch N | NRS score |
| ICEs | Event | Strategy | Description |
| | Discontinuation of intervention or study early prior to Week 16 assessment | Composite variable | Missing data will be imputed using multiple imputation |
| | Lost to follow-up prior to<br>Week 16 or otherwise<br>missing endpoint data at<br>Week 16 assessment | Composite variable | Missing data will be imputed using multiple imputation |
| | Start a protocol prohibited medication/therapy | Treatment policy | Participants will be included in the analysis regardless of the occurrence of the ICE according to the respective endpoint definition. |

Table 10.4.1-1: Definition of Estimands for Primary and Key Secondary Endpoints

| | Missing assessment at<br>Week 16 due to<br>SARS-CoV-2 | While on treatment | Participants will be excluded from the analysis if the Week 16 assessment was not completed due to SARS-CoV-2 |
|---|---|---|---|
| Population-level<br>Summary | Adjusted mean difference b | etween deucrav | vacitinib 6 mg QD and placebo |
| Estimand Attribute | Definition | | |
| Treatment | Deucravacitinib 6 mg QD v | ersus placebo | |
| Population | FAS sub-population | | |
| Variable | s-PGA 0/1 | | |
| ICEs | Event | Strategy | Description |
| | Discontinuation of intervention or study early prior to Week 16 assessment | Composite variable | Participant will be counted as a non-responder |
| | Lost to follow-up prior to<br>Week 16 or otherwise<br>missing endpoint data at<br>Week 16 assessment | Composite variable | Participant will be counted as a non-responder |
| | Start a protocol prohibited medication/therapy | Treatment policy | Participants will be included in the primary analysis regardless of the occurrence of the ICE according to the respective endpoint definition. |
| | Missing assessment at<br>Week 16 due to<br>SARS-CoV-2 | While on treatment | Participants will be excluded from the primary analysis if the Week 16 assessment was not completed due to SARS-CoV-2 |
| Population-level<br>Summary | Odds ratio of achieving s-PGA 0/1 | | |

DLQI, Dermatology Life Quality Index; FAS, Full Analysis Set; ICE, intercurrent event; NRS, Numerical Rating Scale; QD, once daily; SARS-CoV-2, severe acute respiratory syndrome coronavirus 2; s-PGA, static Physician Global Assessment.

# 10.4.2 Primary Endpoint(s)

Table 10.4.2-1: Primary Endpoint

| Primary Endpoint | Description | Timeframe |
|---|---|---|
| DLQI 0/1 | Proportion of participants achieving DLQI score of 0 or 1 | Week 16 |

DLQI, Dermatology Life Quality Index.

Table 10.4.2-2: Summary of Primary Endpoint

| Endpoint | Statistical Analysis Methods |
|---|---|
| DLQI 0/1<br>response rate<br>is defined as a<br>proportion of<br>participants<br>with a DLQI<br>score 0 or 1 | The analysis model for the primary endpoint, DLQI 0/1 (responder/non-responder) at Week 16, will use a stratified CMH test to compare the response rates of deucravacitinib 6 mg QD to placebo using the Week 16 data of the FAS population as well as the FAS subgroup where baseline $s\text{-PGA} \ge 3$ . If expected cell counts are not sufficient for each strata level, then strata levels will be combined for the analysis. The odds ratio (ratio of odds in deucravacitinib 6 mg QD to the odds in placebo group) and the corresponding 2-sided 95% CI will be provided. Estimates of proportions and their 2-sided 95% CIs will be provided. |
| | NRI will be used for the primary efficacy endpoint for participants who discontinue intervention or study prior to Week 16 or who have otherwise missing endpoint data at the specified timepoint. NRI will be the primary method of imputation for the primary efficacy endpoint. |
| | Sensitivity and supportive analyses to be performed for the primary endpoint will be described in the SAP. |

CI, confidence interval; CMH, Cochran-Mantel-Haenszel; DLQI, Dermatology Life Quality Index; NRI, non-responder imputation; QD, once daily; SAP, statistical analysis plan; s-PGA, static Physician Global Assessment.

# 10.4.3 Secondary Endpoint(s)

**Table 10.4.3-1:** Summary of Key Secondary Endpoints

| Endpoint | Statistical Analysis Methods | Time Frame |
|---|---|---|
| ≥ 4-point reduction from baseline in DLQI is defined as a proportion of participants achieving at least a 4-point reduction from baseline in DLQI | The analysis model for $\geq$ 4-point reduction from baseline in DLQI (responder/non-responder) at Week 16, will use stratified CMH tests to compare the response rates of deucravacitinib 6 mg QD to placebo for the FAS population as well as the FAS sub-population where baseline s-PGA $\geq$ 3. If expected cell counts are not sufficient for each strata level, then strata levels will be combined for the analysis. The odds ratio (ratio of odds in deucravacitinib BMS-986165 6 mg QD to the odds in placebo group) and the corresponding 2-sided 95% CI will be provided. Estimates of proportions and their 2-sided 95% CIs will be provided. The NRI method will be applied to the analysis of the binary secondary efficacy endpoint for participants who discontinue early or who have otherwise missing endpoint data at the specified timepoint. | Week 16 |
| Change from<br>baseline in<br>whole-body itch<br>NRS score | The analysis model for the continuous secondary endpoint, change from baseline in whole-body itch NRS at Week 16, will use ANCOVA with intervention . The baseline value will be added into the model as a covariate. Intervention differences based on least-squares means and the corresponding 2-sided 95% CIs will be provided for the difference between deucravacitinib 6 mg QD and placebo for the FAS population as well as the FAS sub-population where baseline s-PGA $\geq 3$ . For the continuous secondary efficacy endpoint, multiple imputation will be used for missing data. | Week 16 |
| Proportion of participants with a s-PGA score of 0 | The analysis model for the secondary endpoint, s-PGA 0/1 (responder/non-responder) at Week 16, will use a stratified CMH) test to compare the response rates of deucravacitinib 6 mg QD to placebo using the | Week 16 |

| Endpoint | Statistical Analysis Methods | Time Frame |
|---|---|---|
| (clear) or 1<br>(almost clear)<br>with at least a<br>2-point<br>reduction from<br>baseline. | Week 16 data of the FAS sub-population where baseline $s-PGA \ge 3$ . If expected cell counts are not sufficient for each strata level, then strata level will be combined for the analysis. The odds ratio (ratio of odds in deucravacitinib 6 mg QD to the odds in placebo group) and the corresponding 2-sided 95% CI will be provided. Estimates of proportions and their 2-sided 95% CIs will be provided. | |
| | The NRI method will be applied to the analysis of the binary secondary efficacy endpoint for participants who discontinue early or who have otherwise missing endpoint data at the specified timepoint. | |

ANCOVA, analysis of covariance; CI, confidence interval; CMH, Cochran-Mantel-Haenszel; DLQI, Dermatology Life Quality Index; FAS, Full Analysis Set; NRI, non-responder imputation; NRS, numerical rating scale; QD, once daily; s-PGA, static Physician Global Assessment.

# 10.4.5 Safety Analysis

Safety data will be analyzed for AEs, SAEs, laboratory parameters, and vital signs. Safety will be summarized using the safety population. Categorical data will be summarized as frequency counts and percentages. Continuous data will be summarized using n, mean, standard deviation, median, minimum, and maximum unless otherwise specified. Safety will be analyzed through Week 16 and then up to end of study.

#### 10.4.5.1 Adverse Events

Treatment-emergent AEs, SAEs, deaths, AEs leading to study intervention discontinuation, will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term.

#### 10.4.5.2 Vital Signs

Vital signs will be summarized as raw, change from baseline, including the maximum post-baseline value. Baseline values are defined as the last non-missing value prior to the first dose of study drug. The number and proportion of participants with vital sign abnormalities will be summarized at each scheduled visit.

# 10.4.5.3 Clinical Laboratory Tests

Laboratory parameters will be summarized as raw, change from baseline, including the maximum post-baseline value. Incidence of abnormal, high, or low values will be summarized. Shift tables will also be provided. Baseline values are defined as the last non-missing value prior to the first dose of study drug. The number and proportion of participants with clinical laboratory abnormalities will be summarized at each scheduled visit.

# 10.4.6 Other Analyses

Not applicable.

Clinical Protocol IM011237 BMS-986165 Deucravacitinib

# 10.5 Interim Analyses

Not applicable.

#### 10.6 Week 16 Primary Analysis

A 16-week primary analysis will occur once all randomized participants have completed their Week 16 visit or have discontinued prior to Week 16. Analyses of the collected efficacy and safety data will be performed. The study participants and investigators will remain blinded to the initial treatment assignment throughout the study. The Sponsor and site facing study team will be unblinded to the individual treatment assignments following the last Week 16 visit.

Additional details of these analyses will be described in the SAP. A final analysis will be performed after all participants complete the final safety follow-up visit at Week 56 or post-discontinuation follow-up visit.

#### 11 REFERENCES

Parisi R, Symmons DP, Griffiths CE, et al. Global epidemiology of psoriasis: a systematic review of incidence and prevalence. J Invest Dermatol. 2013;133(2):377-385.

- <sup>2</sup> Kupetsky EA, Keller M. Psoriasis vulgaris: an evidence-based guide for primary care. J Am Board Fam Med. 2013;26(6):787-801.
- World Health Organization. Global Report on psoriasis. WHO 2016.
- <sup>4</sup> Langely RG, Kruger GG, Griffiths CE. Psoriasis: epidemiology, clinical features, and quality of life. Ann Rheum Dis. 2005;64(Suppl II):ii18-ii23.
- Ouiero R, Tejon P, Alonso S, Coto P. Age at disease onset: a key factor for understanding psoriatic disease. Rheumatology (Oxford). 2014;53(7):1178-1185.
- Merola JF, Qureshi A, Husni ME. Underdiagnosed and undertreated psoriasis: nuances of treating psoriasis affecting the scalp, face, intertriginous areas, genitals, hands, feet, and nails. Dermatol Ther. 2018;31(3):e12589.
- <sup>7</sup> Rapp SR, Feldman SR, Exum ML, et al. Psoriasis causes as much disability as other major medical diseases. J Am Acad Dermatol. 1999;41:401-407.
- de Arruda LH, De Moraes. The impact of psoriasis on quality of life. Br J Dermatol. 2001 Apr;144 Suppl 58:33-36.
- Barbieri JS, Gelfand JM. Patient-Reported Outcome Measures as Complementary Information to Clinician-Reported Outcome Measures in Patients With Psoriasis. JAMA Dermatol. 2021 Oct 1;157(10):1236-1237.
- Golbari NM, van der Walt JM, Blauvelt A et al. Psoriasis severity: commonly used clinical thresholds may not adequately convey patient impact. J Eur Acad Dermatol Venereol. 2021 Feb;35(2):417-421.
- Armstrong AW, Robertson AD, Wu J et al. Undertreatment, treatment trends, and treatment dissatisfaction among patients with psoriasis and psoriatic arthritis in the United States: findings from the National Psoriasis Foundation surveys, 2003-2011. JAMA Dermatol. 2013 Oct;149(10):1180-1185.
- Novartis. Rheumatrex® (methotrexate). United States Prescribing Information. 2016.
- Novartis. Neoral® (cyclosporine). United States Prescribing Information. 2009.
- <sup>14</sup> Celgene. Otezla® (apremilast). United States Prescribing Information. 2017.
- AbbVie. Humira® (adalimumab). United States Prescribing Information. 2017.
- <sup>16</sup> Janssen Biotech. Remicade® (infliximab). United States Prescribing Information. 2013.
- <sup>17</sup> Janssen Biotech. Stelara<sup>®</sup> (ustekinumab). United States Prescribing Information. 2016.
- Novartis. Cosentyx® (secukinumab). United States Prescribing Information. 2015.

- <sup>19</sup> Eli Lilly. Taltz<sup>®</sup> (ixekizumab). United States Prescribing Information. 2017.
- <sup>20</sup> Valeant. Siliq® (brodalumab). United States Prescribing Information. 2017.
- Nestle FO, Kaplan DH, Barker J. Mechanisms of disease: psoriasis. N Engl J Med. 2009;361:496-509.
- <sup>22</sup> Tokarski JS, Zupa-Fernandez A, Tredup JA, et al. Tyrosine kinase 2-mediated signal transduction in T lymphocytes is blocked by pharmacological stabilization of its pseudokinase domain. J Biol Chem. 2015;290:11061-11074.
- Watford WT, Hissong BD, Bream JH, et al. Signaling by IL-12 and IL-23 and the immunoregulatory roles of STAT4. Immunol Rev. 2004;202:139-156.
- Shaw MH, Boyartchuk V, Wong S, et al. A natural mutation in the Tyk2 pseudokinase domain underlies altered susceptibility of B10.Q/J mice to infection and autoimmunity. Proc Natl Acad Sci U S A. 2003:100:11594-11599.
- BMS-986165 Investigator Brochure Version 09. Bristol-Myers Squibb Company; 2022. Document Control No. 930090873.
- <sup>27</sup> Feldman SR, Krueger GG. Psoriasis assessment tools in clinical trials. Ann Rheum Dis. 2005;64:ii65-ii68.
- Fredriksson T, Pettersson U. Severe psoriasis-oral therapy with a new retinoid. Dermatologica. 1978;157(4):238-244.
- Rossiter ND, Chapman P, Haywood IA. How big is a hand? Burns. 1996;22:230-231.
- Long CC, Finlay AY, Averill RW. The rule of hand: 4 hand areas = 2 FTU = 1 g. Arch Dermatol. 1992;128:1129-1130.
- Thomas CL, Finlay AY. The 'handprint' approximates to 1% of the total body surface area whereas the 'palm minus the fingers' does not. Br J Dermatol. 2007;157(5):1080-1081.
- Kragballe K, Menter A, Lebwohl M, et al. Long-term management of scalp psoriasis: perspectives from the international psoriasis council. J Dermatol Treat. 2013;24:188-192.
- Tan EST, Chong W-S, Liang Tey H. Nail psoriasis: a review. Am J Clin Dermatol. 2012;13:375-388.

Clinical Protocol BMS-986165

- Bissonnette R, Pariser DM, Wasel NR, et al. Apremilast, an oral phosphodiesterase-4 inhibitor, in the treatment of palmoplantar psoriasis: Results of a pooled analysis from phase II PSOR- 005 and phase III Efficacy and Safety Trial Evaluating the Effects of Apremilast in Psoriasis (ESTEEM) clinical trials in patients with moderate to severe psoriasis. J Am Acad Dermatol. 2016;75:99-105.
- Lebwohl M, Papp K, Stein Gold L, et al. Trial of roflumilast cream for chronic plaque psoriasis. N Engl J Med. 2020;383(3):229-239.
- Merola J, Bleakman A, Gottlieb A, et al. The Static Physician's Global Assessment of Genitalia: a clinical outcome measure for the severity of genital psoriasis. J Drugs Dermatol. 2017;16(8):793-799.

Protocol Amendment 02

Clinical Protocol IM011237 BMS-986165 Deucravacitinib



<sup>50</sup> Sen PK. Union-intersection principle and constrained statistical inference. Journal of Statistical Planning and Inference. 2007;137(11):3741-3752.

# 12 APPENDICES

# APPENDIX 1 ABBREVIATIONS AND TRADEMARKS

| Term | Definition |
|----------------|---------------------------------|
| <u>AE</u> | adverse event |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| anti-HBc | hepatitis B core antibody |
| anti-HBc total | hepatitis B core antibody total |
| anti-HBs | hepatitis B surface antibody |
| AST | aspartate aminotransferase |
| AxMP | auxiliary medicinal product |
| BID | twice daily |
| BMI | body mass index |
| BMS | Bristol-Myers Squibb Company |
| BP | blood pressure |
| BSA | body surface area |
| CFR | Code of Federal Regulations |
| CI | confidence interval |
| CMH | Cochran-Mantel-Haenszel |
| COVID-19 | coronavirus disease 2019 |
| CRF | Case Report Form |
| CSR | clinical study report |
| CTAg | Clinical Trial Agreement |
| CYP450 | cytochrome P450 |
| DILI | drug-induced liver injury |
| DLQI | Dermatology Life Quality Index |
| DNA | deoxyribonucleic acid |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| e-diary | electronic diary |
| EOT | end of treatment |
| ET | early termination |
| EU | European Union |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |

| Term | Definition |
|---------|--------------------------------------------------------|
| FSH | follicle-stimulating hormone |
| | Tomere summand normone |
| GCP | Good Clinical Practice |
| GIC-SI | Global Impression of Change-Scalp Itch |
| HBsAg | hepatitis B surface antigen |
| HBV | hepatitis B virus |
| hCG | human chorionic gonadotropin |
| HCV | hepatitis C virus |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| HRQoL | health-related quality of life |
| HRT | hormone replacement therapy |
| IB | Investigator's Brochure |
| ICE | intercurrent events |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| ICMJE | International Committee of Medical Journal Editors |
| IEC | Independent Ethics Committee |
| IFN | interferon |
| IL | interleukin |
| IMP | investigational medicinal product |
| IP | investigational product |
| IRT | interactive response technology |
| I-s-PGA | Intertriginous-area static Physician Global Assessment |
| IUS | intrauterine hormone-releasing system |
| JAK | Janus kinase |
| LAM | lactational amenorrhea method |
| MGT | |
| MCT | meaningful change threshold |
| MadDDA | Madical Dictionary for Descriptions Asticities |
| MedDRA | Medical Dictionary for Regulatory Activities |
| n/a | not applicable |
| NIMD | |
| NIMP | non-investigational medicinal product |
| NDI | |
| NRI | non-responder imputation |

| Term | Definition |
|---|---|
| NRS | Numerical Rating Scale |
| PASI | Psoriasis Area and Severity Index |
| 17151 | 1 Sofiasis Area and Severity index |
| PBO | placebo |
| TBO | piaceoo |
| PE | physical examination |
| PGA-F | Physician Global Assessment-Fingernails |
| PGA-G | Physician Global Assessment-Genitals Physician Global Assessment-Genitals |
| TOA-O | Filysician Global Assessment-Genitals |
| | <del> </del> |
| DV | who were a live time. |
| PK | pharmacokinetics |
| PC 4 | 1 1 4 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| pp-PGA | palmoplantar Physician Global Assessment |
| PRO | patient-reported outcome |
| DCO | |
| PSO | psoriasis |
| OD | 1 '1 |
| QD | once daily |
| QoL<br>SAE | quality of life serious adverse event |
| SAP | |
| SARS-CoV-2 | statistical analysis plan severe acute respiratory syndrome coronavirus 2 |
| SARS-COV-2 | severe acute respiratory syndrome coronavirus 2 |
| af DC A | static force Physician Clobal Accessment |
| sf-PGA | static face Physician Global Assessment<br>static Physician Global Assessment |
| s-PGA | |
| s-PGA-G | static Physician Global Assessment Genitalia |
| SSC | Study Steering Committee |
| ss-PGA | scalp-specific Physician Global Assessment |
| STAT | signal transducer and activator of transcription |
| TD | |
| TB | tuberculosis |
| TNF | tumor necrosis factor |
| TSQM | Treatment Satisfaction Questionnaire for Medication |
| TYK2 | tyrosine kinase 2 |
| LILA | 1: '. 6 1 |
| ULN | upper limit of normal |
| US | United States |
| UV | ultraviolet |

| Term | <b>Definition</b> |
|-------|---------------------------------|
| WOCBP | women of childbearing potential |

#### APPENDIX 2 STUDY GOVERNANCE CONSIDERATIONS

The terms "participant" and "subject" refer to a person who has consented to participate in the clinical research study. Typically, the term "participant" is used in the protocol and the term "subject" is used in the Case Report Form (CRF).

#### **REGULATORY AND ETHICAL CONSIDERATIONS**

This study will be conducted in accordance with:

- Consensus ethical principles derived from international guidelines, including the Declaration of Helsinki and Council for International Organizations of Medical Sciences International Ethical Guidelines
- Applicable International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guidelines
- Applicable laws, regulations, and requirements

The study will be conducted in compliance with the protocol. The protocol, any revisions/amendments, and the participant informed consent form (ICF) will receive approval/favorable opinion by Institutional Review Board/Independent Ethics Committee (IRB/IEC), and regulatory authorities according to applicable regulations prior to initiation of the study.

All potential serious breaches must be reported to the Sponsor or designee immediately. A potential serious breach is defined as a Quality Issue (eg, protocol deviation) that is likely to affect, to a significant degree, one or more of the following: (1) the rights, physical safety or mental integrity of 1 or more participants; (2) the scientific value of the clinical study (eg, reliability and robustness of generated data). Items (1) or (2) can be associated with either GCP regulation(s) or study protocol(s).

Personnel involved in conducting this study will be qualified by education, training, and experience to perform their respective tasks.

This study will not use the services of study personnel where sanctions have been invoked or where there has been scientific misconduct or fraud (eg, loss of medical licensure, debarment).

#### INSTITUTIONAL REVIEW BOARD/INDEPENDENT ETHICS COMMITTEE

Before study initiation, the investigator must have written and dated approval/favorable opinion from the IRB/IEC for the protocol, Investigator's Brochure, product labeling information, ICF, participant recruitment materials (eg, advertisements), and any other written information to be provided to participants.

The investigator, Sponsor, or designee should provide the IRB/IEC with reports, updates, and other information (eg, expedited safety reports, amendments, administrative letters) annually, or more frequently, in accordance with regulatory requirements or institution procedures.

Protocol Amendment 02 Date: 25-May-2023 IM011237 Deucravacitinib The investigator is responsible for providing oversight of the conduct of the study at the site and adherence to requirements of the following where applicable:

- ICH guidelines,
- United States Code of Federal Regulations, Title 21, Part 50 (21 CFR 50)
- European Union Directive 2001/20/EC; or
- European Regulation 536/2014 for clinical studies (if applicable),
- European Medical Device Regulation 2017/745 for clinical device research (if applicable),
- the IRB/IEC
- and all other applicable local regulations.

#### COMPLIANCE WITH THE PROTOCOL AND PROTOCOL REVISIONS

The investigator should not implement any deviation or change to the protocol without prior review and documented approval/favorable opinion of an amendment from the IRB/IEC (and, if applicable, also by the local Health Authority), except where necessary to eliminate an immediate hazard(s) to study participants.

If a deviation or change to a protocol is implemented to eliminate an immediate hazard(s) prior to obtaining relevant approval/favorable opinion(s), the deviation or change will be submitted as soon as possible to:

- IRB/IEC
- Regulatory authority(ies), if applicable by local regulations (per national requirements)

Documentation of approval/favorable opinion signed by the chairperson or designee of the IRB(s)/IEC(s) and, if applicable, also by the local Health Authority, must be sent to Bristol-Myers Squibb Company (BMS).

If an amendment substantially alters the study design or increases the potential risk to the participant: (1) the ICF must be revised and submitted to the IRB(s)/IEC(s) for review and approval/favorable opinion; (2) the revised form must be used to obtain consent from participants currently enrolled in the study if they are affected by the amendment; and (3) the new form must be used to obtain consent from new participants prior to enrollment.

#### FINANCIAL DISCLOSURE

Investigators and sub-investigators will provide the Sponsor with sufficient, accurate financial information, in accordance with regulations, to allow the Sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate Health Authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

#### INFORMED CONSENT PROCESS

Investigators must ensure that participants are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which they volunteer to participate.

The Sponsor or designee will provide the investigator with an appropriate sample ICF, which will include all elements required by the ICH GCP, and applicable regulatory requirements. The sample ICF will adhere to the ethical principles that have their origin in the Declaration of Helsinki.

The investigator or his/her representative must:

- Obtain IRB/IEC written approval/favorable opinion of the written ICF and any other information to be provided to the participant prior to the beginning of the study and after any revisions are completed for new information.
- Provide a copy of the ICF and written information about the study in the language in which the participant is proficient prior to clinical study participation. The language must be nontechnical and easily understood.
- Explain the nature of the study to the participant or his/her legally acceptable representative and answer all questions regarding the study.
- Inform participant that his/her participation is voluntary. Participant or his/her legally acceptable representative will be required to sign a statement of informed consent that meets the requirements of 21 CFR 50, local regulations, ICH guidelines, Health Insurance Portability and Accountability Act (HIPAA) requirements, where applicable, and the IRB/IEC or study center.
- Allow time necessary for participant or his/her legally acceptable representative to inquire about the details of the study.
- Obtain an ICF signed and personally dated by the participant or his/her legally acceptable representative and by the person who conducted the informed consent discussion.
- Include a statement in participant's medical record that written informed consent was obtained before participant was enrolled in the study and the date the written consent was obtained. The authorized person obtaining the informed consent must also sign the ICF.
- Re-consent participant to the most current version of the ICF(s) during his/her participation in the study, as applicable.
- Revise the ICF whenever important new information becomes available that is relevant to the participant's consent. The investigator, or a person designated by the investigator, should fully inform the participant or his/her legally acceptable representative of all pertinent aspects of the study and of any new information relevant to the participant's willingness to continue participation in the study. This communication should be documented.

The confidentiality of records that could identify participants must be protected, respecting the privacy and confidentiality rules applicable to regulatory requirements, the participant's signed ICF, and, in the United States (US), the participant's signed HIPAA Authorization.

The ICF must also include a statement that BMS and local and foreign regulatory authorities have direct access to participant records.

In situations where consent cannot be given by participants, their legally acceptable representatives (as per country regulation) are clearly and fully informed about the purpose, potential risks, and other critical issues regarding clinical studies in which the participant volunteers to participate.

If informed consent is initially given by a participant's legally acceptable representative or legal guardian and the participant subsequently becomes capable of making and communicating his or her informed consent during the study, consent must additionally be obtained from the participant.

Participants who are unable to give their written informed consent (eg, due to stroke or participants with severe dementia) may only be enrolled in the study with the consent of a legally acceptable representative. The participant must also be informed about the nature of the study to the extent compatible with his or her understanding, and should this participant become capable, he/she should personally sign and date the ICF as soon as possible. The explicit wish of a participant who is unable to give his or her written consent, but who is capable of forming an opinion and assessing information to refuse participation in, or to be withdrawn from, the clinical study at any time, should be considered by the investigator.

The rights, safety, and well-being of the study participants are the most important considerations and should prevail over interests of science and society.

#### **BMS COMMITMENT TO DIVERSITY IN CLINICAL TRIALS**

The mission of BMS is to transform patients' lives through science by discovering, developing, and delivering innovative medicines that help them prevail over serious diseases.

BMS is committed to doing its part to ensure that patients have a fair and just opportunity to achieve optimal health outcomes.

BMS is working to improve the recruitment of a diverse participant population with the goal that the clinical study becomes more reflective of the real-world population and the people impacted by the diseases studied.

## DATA PROTECTION, DATA PRIVACY, AND DATA SECURITY

BMS collects and processes personal data of study participants, patients, health care providers, and researchers for biopharmaceutical research and development to advance innovative, high-quality medicines that address the medical needs of patients. BMS ensures the privacy, protection, and confidentiality of such personal data to comply with applicable laws. To achieve these goals, BMS has internal policies that indicate measures and controls for processing personal data. BMS adheres to these standards to ensure that collection and processing of personal data are limited and proportionate to the purpose for which BMS collects such personal data. This purpose is clearly and unambiguously notified to the individual at the time of collection of personal data. In the true spirit of science, BMS is dedicated to sharing clinical trial information and data with participants, medical/research communities, the media, policy makers, and the general public. This is done in a manner that safeguards participant privacy and informed consent while respecting the integrity of national regulatory systems. Clinical trial data, health-related research, and

pharmacovigilance activities on key-coded health data transferred by BMS across national borders is done in compliance with the relevant data protection laws in the country and GCP requirements.

BMS protects Personal Information with adequate and appropriate security controls as indicated under the data protection laws. To align with the recommended security standards, BMS has adopted internal security standards and policies to protect personal data at every stage of its processing.

To supplement these standards, BMS enters into Clinical Trial Agreements (CTAgs) with confidentiality obligations to ensure proper handling and protection of personal data by third parties accessing and handling personal data.

BMS takes unauthorized access and disclosure of Personal Information very seriously. BMS has adopted the security standards that include National Institute of Standards and Technology Cybersecurity Framework for studies in the US. BMS aligns with these standards to continuously assess and improve its ability to protect, detect, and respond to cyber attacks and other unauthorized attempts to access personal data. These standards also aid in mitigating possible adverse effects. Furthermore, BMS Information Technology has defined 6 principles to protect our digital resources and information:

- 1. Responsibilities of IT Personnel
- 2. Securing the BMS Digital Infrastructure
- 3. Identity and Access Management
- 4. External Partner Connections
- 5. Cyber Threat Detection and Response
- 6. Internal Cyber Incident Investigation

#### SOURCE DOCUMENTS

Source documents provide evidence for the existence of the participant and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data reported on the CRF or entered in the electronic CRF (eCRF) that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained.

- The investigator may need to request previous medical records or transfer records, depending on the study. Also, current medical records must be available.
- Definitions of what constitutes source data can be found in the source data location list/map or equivalent document.

The investigator is responsible for ensuring that the source data are accurate, legible, contemporaneous, original, and attributable, whether the data are handwritten on paper or entered electronically. If source data are created (first entered), modified, maintained, archived, retrieved, or transmitted electronically via computerized systems (and/or any other kind of electronic devices) as part of regulated clinical study activities, such systems must be compliant with all

applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical records/electronic health records, adverse event (AE) tracking/reporting, protocol-required assessments, and/or drug accountability records.

When paper records from such systems are used in place of an electronic format to perform regulated activities, such paper records should be certified copies. A certified copy consists of a copy of original information that has been verified, as indicated by a dated signature, as an exact copy having all of the same attributes and information as the original.

#### STUDY INTERVENTION RECORDS

Records for study intervention (whether supplied by BMS, its vendors, or the site) must substantiate study intervention integrity and traceability from receipt, preparation, administration, and through destruction or return. Records must be made available for review at the request of BMS/designee or a Health Authority.

| If | Then |
|---|---|
| Supplied by BMS (or its vendors): | Records or logs must comply with applicable regulations and guidelines and should include: • amount received and placed in storage area • amount currently in storage area |
| | • label identification number or batch number |
| | <ul> <li>amount dispensed to and returned by each<br/>participant, including unique participant<br/>identifiers</li> </ul> |
| | • amount transferred to another area/site for dispensing or storage |
| | <ul> <li>nonstudy disposition (eg, lost, wasted)</li> </ul> |
| | • amount destroyed at study site, if applicable |
| | • amount returned to BMS |
| | • retain samples for bioavailability/bioequivalence/biocomparability, if applicable |
| | • dates and initials of person responsible for Investigational Product dispensing/accountability, as per the Delegation of Authority Form |
| Sourced by site and not supplied by BMS or its vendors (examples include Investigational Product sourced from the sites stock or commercial supply or a specialty pharmacy) | The investigator or designee accepts responsibility for documenting traceability and study treatment integrity in accordance with requirements applicable under law and the standard operating procedures/standards of the sourcing pharmacy |

BMS or its designee will provide forms to facilitate inventory control if the investigational site does not have an established system that meets these requirements.

#### **CASE REPORT FORMS**

An investigator is required to prepare and maintain adequate and accurate case histories designed to record all observations and other data pertinent to the investigation on each individual treated or entered as a control in the investigation. Data that are derived from source documents and reported on the CRF must be consistent with the source documents, or the discrepancies must be explained. Additional clinical information may be collected and analyzed in an effort to enhance understanding of product safety. CRFs may be requested for AEs and/or laboratory abnormalities that are reported or identified during the course of the study.

For sites using the Sponsor or designee electronic data capture (EDC) tool, eCRFs will be prepared for all data collection fields except for fields specific to serious adverse events (SAEs) and pregnancy, which will be reported on the electronic SAE form and Pregnancy Surveillance Form, respectively. If the electronic SAE form is not available, a paper SAE form can be used.

The confidentiality of records that could identify participants must be protected, respecting the privacy and confidentiality rules in accordance with the applicable regulatory requirement(s).

The investigator will maintain a signature sheet to document signatures and initials of all persons authorized to make entries and/or corrections on CRFs.

The completed CRF and SAE/pregnancy CRFs must be promptly reviewed, signed, and dated by the investigator or qualified physician who is a sub-investigator and who is delegated this task on the Delegation of Authority Form. Sub-investigators in Japan may not be delegated the CRF approval task. The investigator must retain a copy of the CRFs, including records of the changes and corrections.

Each individual electronically signing eCRFs must meet Sponsor or designee training requirements and must only access the BMS EDC tool using the unique user account provided by the Sponsor or designee. User accounts are not to be shared or reassigned to other individuals.

## **MONITORING**

Monitoring details describing strategy, including definition of study critical data items and processes (eg, risk-based initiatives in operations and quality such as risk management and mitigation strategies and analytical risk-based monitoring), methods, responsibilities, and requirements, including handling of noncompliance issues and monitoring techniques (central, remote, or on-site monitoring) are provided in the monitoring plan.

Representatives of BMS must be allowed to visit all study site locations periodically to assess the data quality and study integrity. On site, they will review study records and directly compare them with source documents, discuss the conduct of the study with the investigator, and verify that the facilities remain acceptable.

Certain CRF pages and/or electronic files may serve as the source documents.

In addition, the study may be evaluated by the Sponsor or designee internal auditors and government inspectors who must be allowed access to CRFs, source documents, other study files, and study facilities. BMS audit reports will be kept confidential.

The investigator must notify BMS promptly of any inspections scheduled by regulatory authorities and promptly forward copies of inspection reports to the Sponsor or designee.

#### **RECORDS RETENTION**

The investigator (or head of the study site in Japan) must retain all study records and source documents for the maximum period required by applicable regulations and guidelines, or institution procedures, or for the period specified by BMS or its designee, whichever is longer. The investigator (or head of the study site in Japan) must contact BMS prior to destroying any records associated with the study.

BMS or its designee will notify the investigator (or head of the study site in Japan) when the study records are no longer needed.

If the investigator withdraws from the study (eg, relocation, retirement), the records shall be transferred to a mutually agreed-upon designee (eg, another investigator, study site, IRB). Notice of such transfer will be given in writing to BMS or its designee.

#### **RETURN OF STUDY TREATMENT**

For this study, study treatments (those supplied by BMS or a vendor or sourced by the investigator), such as partially used study treatment containers, vials, and syringes, may be destroyed on site.

| If | | | Then |
|---|---|---|---|
| Study treatments supplied (including its vendors) | by | BMS | Any unused study interventions supplied by BMS can only be destroyed after being inspected and reconciled by the responsible Study Monitor, unless study treatments containers must be immediately destroyed as required for safety, or to meet local regulations (eg, cytotoxics or biologics). Partially used study interventions and/or empty containers may be destroyed after proper reconciliation and documentation. But unused Investigational Medicinal Product (IMP) must be reconciled by site monitor/Clinical Research Associate prior to destruction. If study treatments will be returned, the return will be arranged by the responsible Study Monitor. |

| If | Then |
|---|---|
| supplied by BMS (or its vendors; eg, study | It is the investigator's or designee's responsibility to dispose of all containers according to the institutional guidelines and procedures. |

It is the investigator's or designee's responsibility to arrange for disposal of study interventions, provided that procedures for proper disposal have been established according to applicable federal, state, local, and institutional guidelines and procedures, and provided that appropriate records of disposal are kept. The following minimal standards must be met:

- On-site disposal practices must not expose humans to risks from the drug.
- On-site disposal practices and procedures are in agreement with applicable laws and regulations, including any special requirements for controlled or hazardous substances.
- Written procedures for on-site disposal are available and followed. The procedures must be filed with the site's standard operating procedures and a copy provided to BMS upon request.
- Records are maintained that allow for traceability of each container, including the date disposed of, quantity disposed, and identification of the person disposing the containers. The method of disposal (eg, incinerator, licensed sanitary landfill, or licensed waste-disposal vendor) must be documented.
- Accountability and disposal records are complete, up to date, and available for the Study Monitor to review throughout the clinical study period.

It is the investigator's or designee's responsibility to arrange for disposal of all empty containers.

If conditions for destruction cannot be met, the responsible Study Monitor will make arrangements for return of study treatments provided by BMS (or its vendors). Destruction of nonstudy treatments sourced by the site, not supplied by BMS, is solely the responsibility of the investigator or designee.

#### STUDY AND SITE CLOSURE

The Sponsor/designee reserves the right to close the study site or to terminate the study at any time for any reason at the sole discretion of the Sponsor. Study sites will be closed upon study completion. A study site is considered closed when all required documents and study supplies have been collected and a study-site closure visit has been performed.

The investigator may initiate study-site closure at any time, provided there is reasonable cause and sufficient notice is given in advance of the intended termination.

- Reasons for the early closure of a study site by the Sponsor or investigator may include, but are not limited to, the following:
- For study termination:
- Discontinuation of further study intervention development
- For site termination:

Clinical Protocol BMS-986165 IM011237 Deucravacitinib

- Failure of the investigator to comply with the protocol, the requirements of the IRB/IEC or local Health Authorities, the Sponsor's procedures, or GCP guidelines
- Inadequate or no recruitment (evaluated after a reasonable amount of time) of participants by the investigator

If the study is prematurely terminated or suspended, the Sponsor shall promptly inform the investigators, the IECs/IRBs, the regulatory authorities, and any contract research organization(s) used in the study of the reason for termination or suspension, as specified by the applicable regulatory requirements. The investigator shall promptly inform the participant and should assure appropriate participant therapy and/or follow-up.

#### **DISSEMINATION OF CLINICAL STUDY DATA**

In order to benefit potential study participants, patients, healthcare providers and researchers, and to help BMS honor its commitments to study participants, BMS will make information about clinical research studies and a summary of their results available to the public as per regulatory and BMS requirements. BMS will post-study information on local, national or regional databases in compliance with national and international standards for disclosure. BMS may also voluntarily disclose information to applicable databases.

In the European Union (EU), the summary of results and summary for laypersons will be submitted within 1 year of the end of trial in EU/European Economic Area and third countries.

#### **CLINICAL STUDY REPORT**

A Signatory Investigator must be selected to sign the clinical study report (CSR).

For each CSR related to this protocol, the following criteria will be used to select the Signatory Investigator:

- External Principal Investigator designated at protocol development
- National Coordinating Investigator
- Study Steering Committee chair or their designee
- Participant recruitment (eg, among the top quartile of enrollers)
- Involvement in study design
- Regional representation (eg, among top quartile of enrollers from a specified region or country)

#### **SCIENTIFIC PUBLICATIONS**

The data collected during this study are confidential and proprietary to the Sponsor or designee. Any publications or abstracts arising from this study must adhere to the publication requirements set forth in the CTAg governing [study site or investigator] participation in the study. These requirements include, but are not limited to, submitting proposed publications to the Sponsor or designee at the earliest practicable time prior to submission or presentation and otherwise within the time period set forth in the CTAg.

Scientific publications (such as abstracts, congress podium presentations and posters, and manuscripts) of the study results will be a collaborative effort between the study Sponsor and the external authors. No public presentation or publication of any interim results may be made by any investigator, sub-investigator, or any other member of the study staff without the prior written consent of the Sponsor.

Authorship of publications at Sponsor is aligned with the criteria of the International Committee of Medical Journal Editors (ICMJE, www.icmje.org). Authorship selection is based upon significant contributions to the study (ie, ICMJE criterion #1). Authors must meet all 4 ICMJE criteria for authorship:

- 1) Substantial intellectual contribution to the conception or design of the work; or the acquisition of data (ie, evaluable participants with quality data), analysis, or interpretation of data for the work (eg, problem solving, advice, evaluation, insights and conclusion); AND
- 2) Drafting the work or revising it critically for important intellectual content; AND
- 3) Final approval of the version to be published; AND
- 4) Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

Those who make the most significant contributions, as defined above, will be considered by BMS for authorship of the primary publication. Sub-investigators will generally not be considered for authorship in the primary publication. Geographic representation will also be considered.

Authors will be listed by order of significant contributions (highest to lowest), with the exception of the last author. Authors in first and last position have provided the most significant contributions to the work.

For secondary analyses and related publications, author list and author order may vary from primary to reflect additional contributions.

# APPENDIX 3 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS: DEFINITIONS AND PROCEDURES FOR RECORDING, EVALUATING, FOLLOW-UP, AND REPORTING

#### ADVERSE EVENTS

#### **Adverse Event Definition:**

An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment that does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.

# **Events Meeting the AE Definition**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or results from other safety assessments (eg, electrocardiograms, radiological scans, vital signs measurements), including those that worsen from baseline, considered clinically significant in the medical and scientific judgement of the investigator. Note that abnormal lab tests or other safety assessments should only be reported as AEs if the final diagnosis is not available. Once the final diagnosis is known, the reported term should be updated to be the diagnosis.
- Exacerbation of a chronic or intermittent pre-existing condition, including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study intervention administration, even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study intervention or a concomitant medication. Overdose, as a verbatim term (as reported by the investigator), should not be reported as an AE/serious adverse event (SAE) unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae and should specify "intentional overdose" as the verbatim term.

#### **Events NOT Meeting the AE Definition**

- Medical or surgical procedure (eg, endoscopy, appendectomy); the condition that leads to the procedure is the AE.
- Situations in which an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).

#### **DEFINITION OF SAE**

If an event is not an AE per definition above, then it cannot be an SAE, even if serious conditions are met.
#### **SERIOUS ADVERSE EVENTS**

## An SAE is defined as any untoward medical occurrence that, at any dose:

Results in death.

Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe).

Requires inpatient hospitalization or causes prolongation of existing hospitalization (see NOTE below).

### NOTE:

The following hospitalizations are not considered SAEs in Bristol-Myers Squibb Company (BMS) clinical studies:

- A visit to the emergency room or other hospital department < 24 hours that does not result in admission (unless considered an important medical or life-threatening event).
- Elective surgery, planned prior to signing consent.
- Admissions as per protocol for a planned medical/surgical procedure.
- Routine health assessment requiring admission for baseline/trending of health status (eg, routine colonoscopy).
- Medical/surgical admission other than to remedy ill health and planned prior to entry into the study. Appropriate documentation is required in these cases.
- Admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention (eg, lack of housing, economic inadequacy, caregiver respite, family circumstances, administrative reason).
- Admission for administration of anticancer therapy in the absence of any other SAEs (applies to oncology protocols).

Results in persistent or significant disability/incapacity.

Is a congenital anomaly/birth defect.

Is an important medical event (defined as a medical event[s] that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgement, may jeopardize the participant or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above). Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm and blood dyscrasias or convulsions that do not result in hospitalization. Potential drug-induced liver injury (DILI) is also considered an important medical event (see Section 9.2.8 for the definition of potential DILI).

Pregnancy and DILI must follow the same transmission timing and processes to BMS as used for SAEs (see Section 9.2.6 for reporting pregnancies).

#### **EVALUATING AES AND SAES**

## **Assessment of Causality**

- The investigator is obligated to assess the relationship between study intervention and each occurrence of each AE/SAE.
- A "reasonable possibility" of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.
- The investigator will use clinical judgement to determine the relationship.
- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study intervention administration, will be considered and investigated.
- The investigator will also consult the Investigator's Brochure and/or product information for marketed products in his/her assessment.
- For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of causality.
- There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the Sponsor. However, it is very important that the investigator always make an assessment of causality for every event before the initial transmission of the SAE data to the Sponsor.
- The investigator may change his/her opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.
- The causality assessment is one of the criteria used when determining regulatory reporting requirements.

## • Assessment of Intensity

The investigator will make an assessment of intensity for each AE and SAE reported during the study and assign it to 1 of the following categories:

- Mild: An event that is easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
- Moderate: An event that causes sufficient discomfort and interferes with normal everyday activities.
- Severe: An event that prevents normal everyday activities. An AE that is assessed as severe should not be confused with an SAE. Severe is a category utilized for rating the intensity of an event, and both AEs and SAEs can be assessed as severe.

An event is defined as "serious" when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, NOT when it is rated as severe.

#### **FOLLOW-UP OF AES AND SAES**

If only limited information is initially available, follow-up reports are required. (Note: Follow-up SAE reports must include the same investigator term[s] initially reported)

If an ongoing SAE changes in its intensity or relationship to study treatment or if new information becomes available, the SAE report must be updated and submitted within 24 hours to BMS (or designee) using the same procedure used for transmitting the initial SAE report.

All SAEs must be followed to resolution or stabilization.

#### REPORTING OF SAES TO SPONSOR OR DESIGNEE

- SAEs, whether related or not related to study treatment, and pregnancies must be reported to BMS (or designee) immediately within 24 hours of awareness of the event.
- SAEs must be recorded on the SAE Report Form.

The required method for SAE data reporting is through the electronic case report form (eCRF).

The paper SAE Report Form is intended only as a back-up option when the electronic data capture system is unavailable/not functioning for transmission of the eCRF to BMS (or designee).

In this case, the paper form is transmitted via email or confirmed facsimile transmission.

When paper forms are used, the original paper forms are to remain on site.

• Pregnancies must be recorded on paper Pregnancy Surveillance Forms and transmitted via email or confirmed facsimile transmission.

SAE Email Address: worldwide.safety@BMS.com

**SAE Facsimile Number:** *Will be provided by local site monitor.* 

**SAE Telephone Contact** (required for SAE and pregnancy reporting): *Will be provided by local site monitor*.

Clinical Protocol IM011237 BMS-986165 Deucravacitinib

# APPENDIX 4 WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION

Appendix 4 provides general information and definitions related to Woman of Childbearing Potential (WOCBP) and methods of contraception that can be applied to most clinical studies. For information specific to this study regarding acceptable contraception requirements for female and male participants, refer to Section 6.1 of the protocol. Only the contraception methods as described in Section 6.1 are acceptable for this study.

#### **DEFINITIONS**

# **Woman of Childbearing Potential**

A woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

# Women in the following categories are not considered WOCBP:

- Premenarchal
- Premenopausal female with 1 of the following:
- Documented hysterectomy
- Documented bilateral salpingectomy
- Documented bilateral oophorectomy

Note: Documentation can come from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

• Postmenopausal female

A postmenopausal state is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle-stimulating hormone (FSH) level > 40 mIU/mL to confirm menopause.

Note: Females treated with hormone replacement therapy (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. Suggested guidelines for the duration of the washout periods for HRT types are presented below. Investigators should use their judgement in checking serum FSH levels.

- 1-week minimum for vaginal hormonal products (rings, creams, gels)
- 4-week minimum for transdermal products
- 8-week minimum for oral products

Other parenteral products may require washout periods as long as 6 months. If the serum FSH level is > 40 mIU/mL at any time during the washout period, the woman can be considered postmenopausal.

# **End of Relevant Systemic Exposure**

End of relevant systemic exposure is the timepoint where the Investigational Medicinal Product (IMP) or any active major metabolites have decreased to a concentration that is no longer considered to be relevant for human teratogenicity or fetotoxicity. This should be evaluated in context of safety margins from the no-observed-adverse-effect level or the time required for 5 half-lives of the IMP to pass.

### **METHODS OF CONTRACEPTION**

Local laws and regulations may require use of alternative and/or additional contraception methods.

# **Highly Effective Contraceptive Methods That Are User Dependent**

Failure rate of < 1% per year when used consistently and correctly.<sup>a</sup>

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation and/or implantation. (This method of contraception can only be used by WOCBP participants in studies where hormonal contraception is permitted by the study protocol)<sup>b</sup>
- Oral (birth control pills)
- Intravaginal (rings)
- Transdermal
- Combined (estrogen-and progestogen-containing) hormonal contraception must begin at least 30 days prior to initiation of study therapy.
- Progestogen-only hormonal contraception associated with inhibition of ovulation. (This method of contraception can only be used by WOCBP participants in studies where hormonal contraception is permitted by the study protocol)<sup>b</sup>
- Oral
- Injectable
- Progestogen-only hormonal contraception must begin at least 30 days prior to initiation of study therapy.

### **Highly Effective Methods That Are User Independent**

- Implantable progestogen-only hormonal contraception associated with inhibition of ovulation and/or implantation. (This method of contraception can only be used by WOCBP participants in studies where hormonal contraception is permitted by the study protocol)b
- Intrauterine device
- Intrauterine hormone-releasing system (IUS). (This method of contraception can only be used by WOCBP participants in studies where hormonal contraception is permitted by the study protocol.)<sup>b,c</sup>
- Bilateral tubal occlusion.
- Vasectomized partner

Having a vasectomized partner is a highly effective contraception method provided that the partner is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

A vasectomy is a highly effective contraception method provided that the participant is the sole male sexual partner of the WOCBP and the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.

#### • Sexual abstinence.

Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.

- Continuous abstinence must begin at least 30 days prior to initiation of study therapy.
- It is not necessary to use any other method of contraception when complete abstinence is elected.
- WOCBP participants who choose complete abstinence must continue to have pregnancy tests, as specified in Section 2.
- Acceptable alternate methods of highly effective contraception must be discussed in the event that the WOCBP participant chooses to forego complete abstinence.
- Periodic abstinence (including, but not limited to, calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM) are not acceptable methods of contraception for this study.

#### NOTES:

- <sup>a</sup> Typical use failure rates may differ from failure rates when contraceptive methods are used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for participants in clinical studies.
- Hormonal contraception may be susceptible to interaction with the study treatment, which may reduce the efficacy of the contraceptive method. Hormonal contraception is permissible only when there is sufficient evidence that the IMP and other study medications will not alter hormonal exposures such that contraception would be ineffective or result in increased exposures that could be potentially hazardous. In this case, alternative methods of contraception should be utilized. For information specific to this study regarding permissibility of hormonal contraception, refer to Section 6.1 INCLUSION CRITERIA and Section 7.7.1 PROHIBITED AND/OR RESTRICTED TREATMENTS of the protocol.
- IUSs are acceptable methods of contraception in the absence of definitive drug interaction studies when hormone exposures from intrauterine devices do not alter contraception effectiveness. For information specific to this study regarding permissibility of hormonal contraception, refer to Section 6.1 INCLUSION CRITERIA and Section 7.7.1 PROHIBITED AND/OR RESTRICTED TREATMENTS of the protocol.

# Less Than Highly Effective Contraceptive Methods That Are User Dependent

Failure rate of > 1% per year when used consistently and correctly

- Male or female condom with or without spermicide. Male and female condoms cannot be used simultaneously
- Diaphragm with spermicide
- Cervical cap with spermicide
- Vaginal sponge with spermicide
- Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mechanism of action. (This method of contraception cannot be used by WOCBP participants in studies where hormonal contraception is prohibited)

### **Unacceptable Methods of Contraception**

- Periodic abstinence (calendar, symptothermal, postovulation methods)
- Withdrawal (coitus interruptus)
- Spermicide only
- LAM

#### **COLLECTION OF PREGNANCY INFORMATION**

Guidance for collection of pregnancy information and outcome of pregnancy on the Pregnancy Surveillance Form is provided in Section 9.2.6 and APPENDIX 3.





# APPENDIX 6 HEPATITIS B VIRUS (HBV) SCREENING

Participants must undergo screening for hepatitis B virus (HBV). At a minimum, this includes testing for HBsAg (hepatitis B surface antigen), anti-HBs (hepatitis B surface antibody), and anti-HBc total (hepatitis B core antibody total):

- Participants who test negative for all HBV screening tests (ie, HBsAg-, anti-HBc-, and anti-HBs-) *are eligible* for this study.
- Participants who test **negative** for surface antigen (HBaAg-) and test positive for core antibody (anti-HBc+) *and* surface antibody (anti-HBs+) *are eligible* for this study.
- Participants who test **positive only** for **surface antibody** (anti-HBs+) **are eligible** for this study.
- Participants who test **positive** for surface antigen (HBsAg+) are NOT eligible for this study, regardless of the results of other hepatitis B tests.
- Participants who test **positive only** for **core antibody** (anti-HBc+) <u>are NOT eligible</u> for this study.

For participants who <u>are not eligible for this study due to HBV test results</u>, consultation with a physician with expertise in the treatment of HBV infection is recommended.

Table 1: Eligibility Based on Hepatitis B Virus Test Results

| | HBV Test Results | | |
|---|---|---|---|
| Action | Hepatitis B Surface<br>Antigen (HBsAg) | Hepatitis B Surface<br>Antibody (anti-HBs) | Hepatitis B Core Antibody<br>Total (anti-HBc total) |
| Include | - | - | - |
| | - | + | - |
| | - | + | + |
| Exclude | + | - or + | - or + |
| | - | - | + |

anti-HBs, hepatitis B surface antibody; anti-HBc, hepatitis B core antibody; HBsAg, hepatitis B surface antigen; HBV, hepatitis B virus.

# APPENDIX 7 PROTOCOL AMENDMENT SUMMARY OF CHANGE HISTORY

# Overall Rationale for Protocol Amendment 01, 21-Nov-2022

The protocol has been revised to add collection at Day 1 (baseline), Week 16, Week 24, and Week 52. The duration that participants will wear the wristwatch increased from 7 days to 14 days prior to each data collection timepoint.

| Summary of Changes for Protocol Amendment 01 | | |
|---|---|---|
| Section Number & Title | Description of Change | Brief Rationale |
| Title Page | Correction of phone number and zip code for address | Updated contact information |
| Schedule of Activities (Table 2-2) | Timepoint of Week -1/Day -7 was changed to Week -2/Day -14 | To reflect current 14-day collection of sleep data prior to Day 1 |
| Schedule of Activities<br>(Table 2-2 and<br>Table 2-3) | | |
| Section 3.1 Study Rationale | The following text was added to reflect FDA approval: "The US Food and Drug Administration (FDA) approved SOTYKTU <sup>TM</sup> (deucravacitinib), a first-in-class, oral, selective, allosteric tyrosine kinase 2 (TYK2) inhibitor, on 09-Sep-2022 for the treatment of adults with moderate-to-severe plaque psoriasis who are candidates for systemic therapy or phototherapy." | To reflect FDA approval of deucravacitinib in the United States |
| Section 3.2.1<br>Clinical Development | The following text was added to reflect FDA approval: "Based on these studies, the US FDA approved SOTYKTU <sup>TM</sup> (deucravacitinib), a first-in-class, oral, selective, allosteric TYK2 inhibitor, on 09-Sep-2022 for the treatment of adults with moderate-to-severe plaque psoriasis who are candidates for systemic therapy or phototherapy." | To reflect FDA approval of deucravacitinib in the United States |
| Section 3.2.1<br>Clinical Development | Updated details regarding completed and ongoing studies. | To include the most up-to-date information in the protocol |

| Summary of Changes for Protocol Amendment 01 | | |
|---|---|---|
| Section Number &<br>Title | Description of Change | Brief Rationale |
| Section 6.3.1<br>Meals and Dietary<br>Restrictions | | |
| Section 9.2.5<br>Pregnancy | The following language was deleted: "Any pregnancy that occurs in a female partner of a male study participant should be reported to Sponsor or designee. In order for Sponsor or designee to collect any pregnancy surveillance information from the female partner, the female partner must sign an ICF for disclosure of this information. Information on this pregnancy will be collected on the Pregnancy Surveillance Form." | To align with current protocol model document language |
| All | Minor formatting and typographical corrections | Minor edits made to improve overall readability, consistency, etc |